Title: A Phase 2a, Multi-center, Double-blind, Placebo-controlled Study Evaluating ABI-H0731 + Entecavir vs Entecavir Alone for the Treatment of Viremic, HBeAg-positive Patients with Chronic Hepatitis B

NCT number: NCT03577171

Date: 18 June 2018



#### CLINICAL RESEARCH PROTOCOL

**PROTOCOL TITLE:** A Phase 2a, Multi-center, Double-blind, Placebo-

controlled Study Evaluating ABI-H0731 + Entecavir vs Entecavir Alone for the Treatment of Viremic, HBeAg-

positive Patients with Chronic Hepatitis B

STUDY NUMBER: ABI-H0731-202

DRUG: ABI-H0731

**REFERENCE NUMBERS:** US IND 136780

**SPONSOR:** Assembly Biosciences

**PROTOCOL:** Amendment 1.0, V2.0, 18 June 2018

Original, V1.0, 15 May 2018

#### **CONFIDENTIAL**

The information contained in this protocol and all other information relevant to Assembly Biosciences are the confidential and proprietary information of Assembly Biosciences and, except as may be required by federal, state, or local laws or regulation, may not be disclosed to others without prior written permission of Assembly Biosciences.

#### CLINICAL PROTOCOL APPROVAL FORM

Protocol Title: A Phase 2a, Multi-center, Double-blind, Placebo-controlled Study Evaluating ABI-H0731 + Entecavir vs Entecavir Alone for the Treatment of Viremic, HBeAg-positive Patients with Chronic Hepatitis B

Study No: ABI-H0731-202 Protocol Date: 18 June 2018

This study protocol was subject to critical review and has been approved by the appropriate protocol review personnel of the Sponsor. The information contained in this protocol is consistent with:

- The current risk-benefit evaluation of the investigational product.
- The ethical and scientific standards governing clinical research that are set out in the current International Council for Harmonisation (ICH) guideline (E6) on Good Clinical Practice (GCP), US Title 21 of the Code of Federal Regulations (CFR) parts 50, 54, 56, and 312, and other applicable local requirements.

The Investigator will be supplied with details of any significant or new findings, including adverse events, relating to treatment with the investigational product.

| Name and Title | Approval Signature | Date |
|----------------|--------------------|------------|
| | | 19June2018 |
| | | 19Jun2018 |

## ABI-H0731-202 PROTOCOL AMENDMENT 1: SUMMARY OF CHANGES

Amendment 1 Dated: 18 June 2018

This document represents the primary changes to Protocol Amendment 1. Changes are either in bold or strikethrough text to note additions or omissions, respectively. For a comprehensive list of the detailed changes made from the Original Protocol to Protocol Amendment 1, refer to the separate redlined (tracked changes) document.

#### 1. CLARIFIED INCLUSION CRITERIA #2 and 6:

Clarified that systemic hormonal birth control (such as oral contraceptive pills or injectable contraceptive depots) are prohibited, whereas, IUDs, including IUDs with hormonal components are allowed. Therefore, Inclusion Criteria #2 has been modified as follows:

• 2. Female subjects must agree to use dual effective birth control methods for the duration of the study and follow-up or be surgically sterile for at least 6 months or at least 2 years postmenopausal, with serum follicle-stimulating hormone (FSH) levels consistent with a postmenopausal status. Effective birth control methods include male or female condom (may not be used together due to increased risk of breakage), vasectomy, intrauterine device (IUD – including IUDs with hormonal components), diaphragm, or cervical cap. Systemic (oral/injectable) hormonal birth control are prohibited. Female subjects must have a negative serum pregnancy test at screening.

Clarified that the Screening laboratory HBV results may be used for the ≥6 month evaluation for the determination of chronic HBV infection as defined in Inclusion #6:

• 6. In good general health except for chronic HBV infection (defined as HBV infection for at least 2 times >6 months documented by − for example − at least two repeated HBsAg positivity and/or history of detectable viral load documented at least two times ≥6 months apart (inclusive of screening), and serum IgM anti-HBV core-related antibody negative at screening

The following sections were updated to reflect these changes:

- Synopsis/Key Eligibility
- Section 5.2/Inclusion Criteria

#### 2. <u>REVISED SECTION 6.6.1/PROHIBITED CONCOMITANT THERAPY</u>

Revised Section 6.6.1/Prohibited Concomitant Therapy to be consistent with the updated Inclusion Criteria #2.

6.6.1 Prohibited Concomitant Therapy

As the potential for drug-drug interactions between ABI-H0731 and other compounds has not yet been fully evaluated, consumption of grapefruit/grapefruit juice is forbidden. **Systemic** 

(oral, injectable, or implanted) hormonal birth control is not permitted as an acceptable means of birth control for female subjects of child bearing potential. Additional prescription medication use is discouraged, unless required for an emergent medical need occurring during the course of the study....

## 3. <u>REVISED SECTION 4.6.1: SUBJECTS WITH ALANINE AMINOTRANSFERASE ELEVATIONS</u>

Revised Section 4.6.1/Subjects with Alanine Aminotransferase Elevations per the request of a regulatory agency:

Subjects experiencing ALT elevations ≥2×Baseline **or on-treatment nadir** and >2×upper limit of normal (ULN) during study treatment or during post-treatment follow-up will be closely monitored. The following guidance is offered for management of study subjects with ALT elevations or biochemical evidence of deteriorating declining hepatic function—("possible decompensation"):

- ALT flare on treatment
  - All subjects with an ALT flare on treatment, defined as ALT>2×Baseline or ontreatment nadir and ≥10×ULN, should have the ALT findings confirmed within 3 days of receipt of the original results....
    - If an intercurrent cause is determined to be causal, the intercurrent cause should be treated as deemed medically appropriate by the Study Investigatortreating physician.
    - In the absence of evidence of possible decompensation declining hepatic function, and in the absence of contraindications, subjects with an ALT flare may continue on study under close observation, with unscheduled visits as deemed necessary by the Study Investigator.
      - o If ALT is rising at the confirmatory visit, subjects should return for an unscheduled visit every 2-5 days until the ALT elevation has stabilized. Subsequently, sSubjects whose ALT has stabilized should continue to be monitored at least weekly (or more frequently as deemed necessary by the treating physician) until ALT values return to normal or baseline levels.
    - Subjects with ALT "flares" or ALT elevations without declining hepatic function or contraindications should stop study drug if the ALT remains persistently elevated for > two weeks in the absence of decreasing HBV DNA (if detectable), and/or HBV RNA, and/or viral antigen (HBeAg or HBsAg).
  - Declining hepatic function during treatment
    - o Subjects with confirmed biochemical evidence of deteriorating declining hepatic function, ie, a direct bilirubin increase to ≥2×Baseline and ≥2×ULN, an albumin

decline ≥0.5 g/dL, INR >2×Baseline and >2×ULN, with an associated ALT elevation ≥2×Baseline and >2×ULN, should be discontinued from study treatment. **Declining** hepatic function is defined as:

- ALT elevation ≥2 × Baseline or nadir and >2×ULN AND
  - Direct bilirubin increase to  $\ge 2 \times Baseline$  and  $\ge 2 \times ULN$  OR
  - o An albumin decline ≥0.5 g/dL OR INR >2×Baseline OR
  - Symptoms of liver inflammation (fatigue, weakness, lack of appetite, nausea, vomiting, jaundice or discolored feces)
- Subjects with evidence of declining hepatic function should return for an unscheduled visit every 2-5 days until the relevant laboratory values stabilize. Subjects whose hepatic function has stabilized should continue to be monitored weekly (or more frequently if deemed necessary by the treating physician) until the relevant laboratory values return to normal or baseline.
- Post-treatment ALT "flare" or ALT elevation with possible decompensation declining hepatic function
  - o For subjects who elect not to enroll in the open-label, extension study ABI-H0731-211, risk of post-treatment flare is mitigated by advising subject to continue on ETV for CHB. Any subject with a post-treatment ALT elevation meeting the ALT "flare" definition (described above)(ALT ≥2×Baseline and ≥10×ULN while on treatment with a regulatory-approved HBV antiviral agent should return for an unscheduled visit every 2-5 days until the relevant laboratory values stabilize. Subjects whose hepatic function has stabilized should continue to be monitored weekly (or more frequently as deemed necessary by the treating physician) until the relevant laboratory values return to normal or baseline levels. Subsequently, subjects should-continue to be followed on their regular study visit schedule, with the addition of any unscheduled visits the Principal Investigator believes are merited for the safety and well-being of the subject.

All subjects with declining hepatic function or ALT flare (on or off treatment) should continue to be followed on their regular study visit schedule, with the addition of unscheduled visits **as described abovedeemed warranted by the Principal Investigator**. If the post-treatment ALT flare has not substantially resolved by the last study follow-up visit, subjects should continue to return to clinic....

If 2 or more subjects meet these LFT flare management criteria, the US FDA and other relevant regulatory agencies will be notified.

## 4. REVISED SECTIONS TO BE CONSISTENT WITH SECTION 4.6.1/ SUBJECTS WITH ALANINE AMINOTRANSFERASE ELEVATIONS

Various sections of the protocol were revised to be consistent with the definitions of ALT flare and declining hepatic function per section 4.6.1/Subjects with Alanine Aminotransferase Elevations.

• 7.2.1 Discontinuation from Treatment

- ... In this study, subjects will be closely monitored for any evidence of worsening hepatic function or evidence of dermatologic adverse events. Subjects with post-Baseline ALT elevations of 2-fold or higher will be closely monitored. Study treatment will be discontinued in any subjects with **confirmed** evidence of declining hepatic function during treatment, ie, bilirubin elevations to >2×ULN or confirmed 0.5 g/dL declines in albumin, with an associated ALT elevation, or increase in INR >2×Baseline and >2×ULN (Section 4.6.1)...
- Appendix II/Adverse Event Intensity Grading was modified as follows:
  - o The following Laboratory Values: Chemistries were added:

| Parameter | Grade 1 Mild | Grade 2 Moderate | Grade 3 Severe | Grade 4 Potentially Life- Threatening |
|---|---|---|---|---|
| Albumin, Low | 3.0 to < LLN | ≥ 2.0 to < 3.0 | < 2.0 | NA |
| (g/dL; g/L) | 30 to < LLN | $\geq 20 \text{ to} < 30$ | < 20 | |
| Alkaline Phosphatase, High | 1.25 to < 2.5 x ULN | 2.5 to < 5.0 x ULN | 5.0 to < 10.0 x ULN | $\geq$ 10.0 x ULN |
| Alkalosis | NA | pH > ULN to ≤ 7.5 | pH > 7.5 without life-<br>threatening<br>consequences | pH > 7.5 with<br>life-threatening<br>consequences |
| ALT or SGPT, High Report only one | 1.25 to < 2.5 x ULN | 2.5 to < 5.0 x ULN | 5.0 to < 10.0 x ULN | ≥ 10.0 x ULN |
| Amylase (Pancreatic) or<br>Amylase (Total), High<br>Report only one | 1.1 to <1.5×ULN | 1.5 to <3.0×ULN | 3.0 to <5.0×ULN | ≥5.0×ULN |
| AST or SGOT, High Report only one | 1.25 to < 2.5 x ULN | 2.5 to < 5.0 x ULN | 5.0 to < 10.0 x ULN | ≥ 10.0 x ULN |
| Bilirubin<br>Direct Bilirubin, High | NA | NA | > ULN with other<br>signs and symptoms of<br>hepatotoxicity <del>.</del> | > ULN with life-<br>threatening<br>consequences<br>(e.g., signs and<br>symptoms of<br>liver failure) |

#### 5. CORRECTED AND REVISED THE SCHEDULE OF ASSESSMENTS (TABLE 1)

The following corrections and revisions were made to the Schedule of Assessments/Table 1:

- Informed Consent(s)
  - o Footnote d was revised for clarity as follows:
    - d. Study specific including optional PG consent. PG sample collection requires documentation of completed PG consent. Subjects who elect to roll over onto the open-label extension study will be required to sign a separate consent at Week 24.
  - O Added to the Table that this assessment is to be performed at Week 24 and added Footnote l. To clarify, subjects are to sign a separate consent form specific to openlabel extension study (ABI-H0731-211) if they choose to participate in that study. Footnote l has been added to the Schedule of Assessments as follows:

- 1. Subjects who elect to roll over onto the open-label extension study will be required to sign a separate consent at Week 24.
- Study Drug Accountability was revised to <u>Study-Drug accountability</u> to clarify reference to combination therapy of ETV ± ABI-H0731
- Study Drug Dispensation was revised to Study Drug dispensation to clarify reference to combination therapy of ETV ± ABI-H0731
- In-clinic dosing: study drug
  - o The line was revised to In-clinic dosing: study drug ABI-H0731/placebo
  - Footnote k was revised for clarity:
    - k. At non-PK collection visits, ETV may be taken outside of the clinic visit pPer package insert instructions for dosing. Of note, ETV is recommended to be dosed 2 hours before or after eating. If subjects are not able to remain in clinic for ETV dosing, then ETV may be dosed following their clinic visits and subjects should be reminded to record the dosing time within their dosing diary. Subjects should not time of dosing and provide this information to the site at the earliest opportunity.
- Footnote c was revised to be consistent with the definition of ALT flare:
  - c. Any subjects with rash or ALT flare (defined in section 4.6-as ALT≥2×Baseline [or 2× on-treatment nadir] and ≥10×ULN) should return to the clinic for an unscheduled visit as soon as possible, ideally within 3 days

#### 6. ADMINISTRATIVE CHANGES

The following changes were made throughout the protocol:

- Table 3/Pharmacokinetic Sample Collection was revised for clarity.
  - The Time Relative to Study Drug Administration for the Day 1 pre-dose and the Study Weeks 2, 4, 12, 24 pre-dose samples were changed from "Immediately Before" to "Immediately Before".
- The Protocol Synopsis was updated to be consistent with the revisions made to the body of the protocol per Amendment 1
- Minor changes have been throughout the document made to improve clarity and consistency between sections. Misspellings and typographical errors were corrected and the document was formatted so that section numbering would be consistent.

#### ABI-H0731-202

# A PHASE 2A, MULTI-CENTER, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY EVALUATING ABI-H0731+ ENTECAVIR VERSUS ENTECAVIR ALONE FOR THE TREATMENT OF VIREMIC, HBEAG-POSITIVE PATIENTS WITH CHRONIC HEPATITIS B

#### INVESTIGATOR STATEMENT

I have read the protocol, including all appendices, and I agree that it contains all of the necessary information for me and my staff to conduct this study as described. I will conduct this study as described herein, in accordance with Good Clinical Practice (GCP) as set out in the current International Council for Harmonisation (ICH) guidelines (E6) and other applicable national or local requirements, and will make a reasonable effort to complete the study within the time designated.

I will provide all study personnel under my supervision copies of the protocol and any amendments, and access to all information provided by Assembly Biosciences or specified designees. I will discuss the material with them to ensure that they are fully informed about Assembly Biosciences and the study.

| Principal Investigator Name (printed) | Signature |
|---------------------------------------|-------------|
| Date | Site Number |

Please keep the original, signed copy of this Investigator signature page in your records and email a copy to your Clinical Research Associate.

#### 1 SYNOPSIS

Protocol ABI-H0731-202 Number:

Title: A Phase 2a, Multi-center, Double-blind, Placebo-controlled Study Evaluating ABI-

H0731 + Entecavir versus Entecavir Alone for the Treatment of Viremic, HBeAg-

positive Patients with Chronic Hepatitis B

Phase: 2a

Number of Subjects:

Approximately 24

**Study Duration:** Up to 45 days for screening, 6 months treatment, and 3 months follow-up

**Rationale:** Chronic hepatitis B infection (CHB) is a major global cause of severe liver morbidity and

liver-related mortality. ABI-H0731 is a direct acting antiviral targeting the hepatitis B virus (HBV) core protein. It is anticipated that ABI-H0731 in combination with entecavir (ETV), a standard of care (SOC) nucleos(t)ide analogue (NUC) therapy, will be safe and increase the functional cure rate for treatment-naïve patients with CHB. This study will explore the safety of combination therapy, as well as its potential for enhanced anti-viral efficacy as measured by the improvement in serum viral DNA reductions, effect on serum biomarkers of functional cures: quantitative and qualitative reduction in the viral antigens hepatitis B "e" antigen (HBeAg) and hepatitis B surface antigen (HBsAg), and reduction in circulating

HBV RNA.

Target Male or female HBeAg-positive treatment-naïve subjects with CHB, age 18 to 70 years,

**Population:** with no evidence of cirrhosis or end-stage liver disease.

**Test Product:** Active treatment subjects will receive ABI-H0731 300 mg, administered orally, once daily,

as three 100-mg tablets in addition to ETV therapy.

**Reference** Placebo subjects will receive placebo (matching ABI-H0731 100-mg tablets), administered

**Product:** orally, once daily, as three tablets in addition to ETV therapy.

Study Design: This is a Phase 2a, multi-center, randomized, double-blind, placebo-controlled study

evaluating the safety, efficacy, pharmacokinetics (PK), and pharmacodynamics of ABI-H0731 in combination with ETV in treatment-naïve subjects with HBeAg-positive CHB virus infection. Subjects will be randomized 1:1 to receive investigational agent (ABI-H0731 or matching placebo) as add-on therapy to ETV for up to 6 months. Efficacy, safety, and PK will be assessed during the 6-month treatment period. At the end of the study treatment period, subjects will have the option to roll over into an optional, open-label, extension study of ABI-H0731 + SOC NUC (protocol ABI-H0731-211) or continue

receiving ETV therapy and stop treatment with ABI-H0731/placebo.

#### **Objectives:**

#### **Primary:**

• To evaluate the potential for ABI-H0731 to increase the rapidity of HBV DNA loss in HBeAg-positive CHB subjects by initiating treatment with ABI-H0731 + ETV in subjects who are not yet on treatment for CHB, as measured by timing and magnitude of change in serum HBV DNA from Baseline

#### **Secondary:**

- To evaluate the safety and tolerability of ABI-H0731 when added to ETV therapy as initial therapy for HBeAg-positive CHB subjects
- To confirm a lack of drug-drug interactions between ETV and ABI-H0731
- To evaluate the potential for emergence of resistance, if any, to ABI-H0731 in combination with ETV therapy

#### **Exploratory:**

- To evaluate the kinetics of and absolute changes from Baseline in biomarkers of transcriptionally active cccDNA (HBeAg and HBsAg)
- To evaluate the kinetics of and absolute changes from Baseline in circulating viral RNA
- To assess the relationship between exploratory viral biomarkers such as changes in viral RNA and hepatitis B core-related antigen (HBCrAg) and outcome
- To explore the PK of ABI-H0731
- For subjects who provide an optional pharmacogenomic sample, to evaluate the potential contribution of host genomics to outcomes

#### Primary Endpoint:

The primary efficacy endpoint will be:

• Change in mean log<sub>10</sub> HBV DNA from Baseline (Day 1) to Week 12 or Week 24 on ABI-H0731 + ETV as compared to placebo + ETV

## Secondary Endpoints:

#### Secondary endpoints will be:

- Number of subjects with adverse events, premature discontinuations, abnormal safety laboratory results, electrocardiogram (ECG), or vital signs
- Subjects with abnormal alanine aminotransferase (ALT) at Baseline who have normal ALT at Week 24 on ABI-H0731 + ETV as compared to placebo + ETV
- Percent of subjects with a decline in viral DNA to below limit of quantitation (LOQ; on ABI-H0731 + ETV as compared to placebo + ETV) at end of treatment
- Median time to viral suppression, defined as HBV DNA <20 IU/mL, on ABI-H0731 + ETV as compared to placebo + ETV
- Emergence of resistant HBV variants, if any
- Drug concentrations:
  - Trough levels and (in subjects where optional post-dose samples are available) trough to peak ratios of ABI-H0731 on ABI-H0731 + ETV therapy
  - O Trough levels and (in subjects where optional post-dose samples are available) trough to peak ratios of ETV on ABI-H0731 + ETV therapy as compared with placebo + ETV therapy

## Exploratory Endpoints:

Exploratory endpoints will include:

- Quantitative changes in serum viral antigen (HBsAg or HBeAg, and HBCrAg) on ABI-H0731 + ETV as compared with placebo + ETV, at each time point
- Subjects with loss (defined as below LOQ) or decline in HBsAg or HBeAg (<0.5 log<sub>10</sub>, ≥0.5 to 1.0 log<sub>10</sub>, or >1.0 log<sub>10</sub> decrease in viral antigen) on ABI-H0731 + ETV as compared with placebo + ETV at end of treatment and end of follow-up
- Subjects with HBsAg seroconversion (loss of HBsAg and appearance of HBs antibody) or HBeAg seroconversion (loss of HBeAg and appearance of HBe antibody) on ABI-H0731 + ETV as compared with placebo + ETV
- Quantitative changes from Baseline in mean log<sub>10</sub> viral RNA, on ABI-H0731 + ETV, as compared with placebo + ETV, at each time point
- Subjects whose HBV DNA achieves "target not detected" on ABI-H0731 + ETV as compared with placebo + ETV
- For subjects who do NOT rollover onto the optional, extension study, ABI-H0731-211:
  - Subjects with suppression of detectable serum HBV RNA on treatment whose RNA rebounds after discontinuing treatment with ABI-H0731 + ETV as compared with placebo + ETV therapy
  - Subjects with changes in HBsAg or HBeAg from Baseline whose viral antigen rebounds after discontinuing investigational treatment with ABI-H0731 + ETV as compared with placebo + ETV
  - Subjects with HBsAg or HBeAg loss at Week 24 that is maintained through end of Follow-up (Week 36) after discontinuing investigational treatment with ABI-H0731 + ETV as compared with placebo + ETV
- If differences are seen in outcomes/adverse events between racial or ethnic groups: Pharmacogenomics correlation with clinical outcomes subjects who provide optional informed consent

## Statistical Methods:

As a proof-of-concept trial, there are no statistical hypotheses, per se, regarding treatment effects in this study. Rather, displays and comparisons of study results, regarding doserelated safety, efficacy, and PK profiles among the treatment groups, will primarily utilize descriptive statistics, as noted below.

The primary comparison for the primary variable will be made using a two-sided, two-sample t-test for mean differences with alpha=0.05.

Secondary and exploratory endpoints will be analyzed descriptively. All secondary and exploratory efficacy endpoints will be summarized.

For continuous variables, such as observed and change from Baseline HBV DNA values at each timepoint, descriptive statistics will be used and will include the number, mean, standard deviation, median, minimum, maximum, and interquartile range and, where appropriate, a 95% confidence interval (CI).

For categorical variables, such as subjects with a 1 log<sub>10</sub> drop in serum HBsAg titers from Baseline and subjects with HBeAg (or HBsAg) loss and seroconversion, descriptive statistics will include number and percent who meet the endpoint criteria.

Kaplan-Meier methods will be used to evaluate time to HBsAg and HBeAg loss (ie, antigen levels less than LOQ), and the treatment groups will be compared using log-rank tests.

Cox proportional hazards regression models will be used to identify baseline factors associated with HBsAg and HBeAg loss rates, as defined in the statistical analysis plan.

#### Key Eligibility:

#### **Inclusion Criteria**

Subjects must meet inclusion criteria in order to be eligible for enrollment.

- 1. Male or female between ages 18 and 70 years (inclusive)
- 2. Female subjects must agree to use dual effective birth control methods for the duration of the study and follow-up or be surgically sterile for at least 6 months or at least 2 years post-menopausal, with serum follicle-stimulating hormone (FSH) levels consistent with a post-menopausal status. Effective birth control methods include male or female condom (may not be used together due to increased risk of breakage), vasectomy, intrauterine device (IUD), diaphragm, or cervical cap. Systemic (oral/injectable) hormonal birth control are prohibited. Female subjects must have a negative serum pregnancy test at screening
- 3. All heterosexually active male subjects must agree to use dual effective birth control methods for the duration of the study and follow-up. Effective birth control methods include male or female condom (may not be used together due to increased risk of breakage), vasectomy, hormone-based, IUD, diaphragm, or cervical cap
- 4. Body mass index (BMI) 18 to 36 kg/m<sup>2</sup> and a minimum body weight of 45 kg (inclusive)
- 5. Agreement to adhere to Lifestyle Considerations (including abstaining from alcohol abuse [defined as alcohol consumption exceeding 2 standard drinks per day on average (1 standard drink = 10 grams of alcohol)] and the use of illicit substances, herbal or other substances, or unnecessary over-the-counter medications; see Protocol Section 5.4) throughout study duration
- 6. In good general health except for chronic HBV infection (defined as HBV infection for at least 6 months documented by for example by two repeated HBsAg positivity and/or detectable viral load documented at least two times ≥6 months apart (inclusive of screening), and serum IgM anti-HBV core-related antibody negative at screening
- 7. HBV viral load ≥2×10<sup>5</sup> IU/mL
- 8. HBeAg-positive at screening
- 9. HBsAg >1000 IU/mL at screening
- 10. Liver biopsy results of
  - o Metavir F0-F2 (absence of bridging fibrosis or cirrhosis) within 1 year of screening

#### OR

o Fasting FibroScan ≤8 kPa within 3 months of screening (including screening visit) or other Sponsor-approved hepatic imaging study (hepatic magnetic resonance imaging [MRI], or hepatic ultrasound by a ultrasongrapher with expertise in

evaluation of liver fibrosis) within 6 months of screening indicating lack of cirrhosis or advanced liver disease (F0-F2 or equivalent).

Subjects with an ambiguous non-invasive result, eg, a fasting FibroScan >8 kPa and  $\le$ 10 kPa are excluded unless a biopsy within the 12 months before first visit confirms the absence of bridging fibrosis and cirrhosis. Subjects with a FibroScan >10 kPa are excluded

- 11. Have the ability to take oral medication and be willing to adhere to the ABI-H0731-202 regimen in the opinion of the Investigator
- 12. Willing and able to provide informed consent

#### **Exclusion Criteria**

Subjects who meet exclusion criteria will not be eligible for enrollment.

- 1. Co-infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV), hepatitis E virus (HEV), or hepatitis D virus (HDV)
- 2. History or evidence of hepatic decompensation (including gastrointestinal bleeding or esophageal varices) at any time prior to or at time of screening
- 3. Subject is febrile (temperature >37.5°C) at screening
- 4. Clinically significant cardiac or pulmonary disease, chronic or recurrent renal or urinary tract disease, liver disease other than HBV, endocrine disorder, autoimmune disorder, diabetes mellitus requiring treatment with insulin or hypoglycemic agents, neuromuscular, musculoskeletal, or mucocutaneous conditions requiring frequent treatment, seizure disorders requiring treatment, or other medical conditions requiring frequent medical management or pharmacologic or surgical treatment that in the opinion of the Investigator or the Sponsor makes the subject unsuitable for the study
- 5. Any prior treatment with lamivudine or telbivudine, previous treatment with an investigational agent for HBV other than ABI-H0731; or any other SOC treatment for >4 weeks
- 6. Participation in another clinical trial of a drug or device whereby the last investigational drug/device administration is within 60 days or five half-lives prior to the first study drug administration, whichever is longer
- 7. History of persistent ethanol abuse (alcohol consumption exceeding 2 standard drinks per day on average [1 standard drink = 10 grams of alcohol]) or illicit drug abuse within 3 years before screening
- 8. Females who are lactating or pregnant or wish to become pregnant
- 9. History of hepatocellular carcinoma (HCC)
- 10. A history of malignancy other than HCC unless the subject's malignancy has been in complete remission off chemotherapy and without additional medical or surgical interventions during the 3 years before screening
- 11. Exclusionary laboratory results
  - a. Platelet count <100,000/mm<sup>3</sup>
  - b. Albumin < lower limit of normal (LLN)

- c. Total bilirubin >1.2×upper limit of normal (ULN) unless known Gilbert syndrome; subjects with Gilbert syndrome are eligible if direct bilirubin is within normal limits
- d. Direct bilirubin >1.2×ULN
- e. ALT >10×ULN at screening
- f. Serum alpha fetoprotein (AFP) ≥100 ng/mL. If AFP at screening is >ULN but <100 ng/mL, subject is eligible if a hepatic imaging study prior to initiation of study drug reveals no lesions suspicious of possible HCC
- g. Prothrombin time: International Normalized Ratio (INR) >1.5×ULN
- h. Glomerular filtration rate (GFR) <60 mL/min/1.73 m<sup>2</sup> by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation [Levey 2009]
- i. Serum hemoglobin A1c (HbA1c) >8%
- j. Any other laboratory abnormality deemed clinically significant by the Sponsor or the Investigator

### **TABLE OF CONTENTS**

| 1 | SYNOPSIS | 9 |
|---|---|---|
| 2 | INTRODUCTION AND RATIONALE | 21 |
| 2.1 | Study Rationale | 21 |
| 2.2 | Background | 21 |
| <b>2.2.</b> 1 | 1 Chronic Hepatitis B Virus | 21 |
| 2.2.2 | 2 Hepatitis B Virus Biology and Rationale for Hepatitis B Virus Core Protein | 1 |
| | Allosteric Modifiers (CpAMs) | |
| 2.2.3 | Summary of Nonclinical Pharmacology and Toxicology | 24 |
| 2.2.4 | | |
| 2.3 | Risk/Benefit Assessment | <b> 26</b> |
| <b>2.3.</b> 1 | 1 Known and Potential Risks of ABI-H0731 | <b> 26</b> |
| 2.3.2 | 2 Known and Potential Benefits of ABI-H0731 | 27 |
| 2.3.3 | Assessment of Potential Risks and Benefits | 28 |
| 3 | STUDY OBJECTIVES AND ENDPOINTS | <b>29</b> |
| 3.1 | Objectives | <b>29</b> |
| <b>3.1.</b> 1 | Primary Objective | <b>29</b> |
| 3.1.2 | Secondary Objectives | <b>29</b> |
| 3.1.3 | Exploratory Objectives | 29 |
| 3.2 | Study Endpoints | |
| <b>3.2.</b> 1 | Primary Endpoint | <b>29</b> |
| 3.2.2 | Secondary Endpoints | 30 |
| <b>3.2.</b> 3 | 3 Exploratory Endpoints | 30 |
| 4 | STUDY PLAN | 32 |
| 4.1 | Study Design | 32 |
| 4.2 | Scientific Rationale | 32 |
| 4.3 | Dose Justification | 33 |
| 4.4 | Study Drug Resistance Monitoring | 33 |
| 4.5 | End of Study Definition | |
| 4.6 | Management of Toxicities | |
| <b>4.6.</b> 1 | | |
| 4.6.2 | 2 Subjects with Rash | 35 |
| <b>4.7</b> | Study Schematic | 36 |
| 4.8 | Schedule of Assessments | |
| 5 | POPULATION | |
| <b>5.1</b> | Number of Subjects | |
| <b>5.2</b> | Inclusion Criteria | 40 |
| <b>5.3</b> | Exclusion Criteria | |
| <b>5.4</b> | Lifestyle Considerations | |
| <b>5.5</b> | Screen Failures | |
| <b>5.6</b> | Strategies for Recruitment and Retention | |
| 6 | STUDY DRUG | |
| 6.1 | Description | 44 |

| 6.1.1 | Formulation | . 44 |
|--------------|------------------------------------------------|------|
| <b>6.1.2</b> | Storage | 44 |
| <b>6.2</b> | Packaging and Shipment | 45 |
| 6.3 | Dose and Administration | 45 |
| 6.3.1 | Dosing in the Study | 45 |
| 6.3.2 | Preparation | 45 |
| 6.3.3 | Blinding | 45 |
| 6.4 | Accountability | 45 |
| 6.5 | Compliance | 46 |
| 6.6 | Concomitant Therapy | 46 |
| 6.6.1 | Prohibited Concomitant Therapy | 46 |
| 6.6.2 | Other Medications and Treatments | |
| <b>7 S</b> 7 | FUDY CONDUCT | 47 |
| <b>7.1</b> | Study Procedures by Time Point | 47 |
| <b>7.2</b> | Discontinuation | 47 |
| <b>7.2.1</b> | Discontinuation from Treatment | 47 |
| 7.2.2 | Discontinuation from Study | 47 |
| 8 D | ESCRIPTION OF STUDY PROCEDURES | 48 |
| 8.1 | Efficacy Assessments | 48 |
| 8.1.1 | Primary Efficacy Assessment | 48 |
| 8.1.2 | Secondary and Exploratory Efficacy Assessments | |
| 8.2 | Safety Assessments. | |
| 8.2.1 | Clinical Laboratory Tests | 49 |
| 8.2.2 | Other Safety Assessments | |
| 8.3 | Pharmacokinetic Assessments | 50 |
| 8.4 | Other Assessments | 50 |
| 8.5 | Protocol Deviations | 51 |
| 9 A | DVERSE EVENTS | 52 |
| 9.1 | Documenting Adverse Events | 52 |
| 9.2 | Assessment of Intensity | |
| 9.3 | Assessment of Causality | 53 |
| 9.4 | Expectedness | 53 |
| 9.5 | Adverse Events of Special Interest | 53 |
| 9.6 | Clinical Laboratory Changes | 53 |
| <b>9.7</b> | Adverse Event Follow-up | 54 |
| 9.8 | Pregnancy | 54 |
| 10 SI | ERIOUS ADVERSE EVENT | 55 |
| 10.1 | Definition of Serious Adverse Event | 55 |
| 10.2 | Reporting Serious Adverse Events | 56 |
| 10.3 | Overdose | |
| 11 S | FATISTICS | |
| 11.1 | Statistical Hypotheses | 58 |
| 11.2 | Sample Size | |
| 11.3 | Analysis Populations | |
| 11.4 | Statistical Methods | 59 |

| 11.4.1 | General Considerations | <b>59</b> |
|---|---|---|
| 11.4.2 | | |
| 11.4.3 | Secondary and Exploratory Endpoint(s) | <b>59</b> |
| 11.4.4 | Pharmacokinetic Endpoints and Analyses | |
| 11.4.5 | Analysis of Safety | 60 |
| 11.4.6 | Demographic and Baseline Characteristics | |
| 11.5 | Interim Analysis | 61 |
| 11.6 | Exploratory Analyses | 61 |
| 12 E | THICS AND RESPONSIBILITIES | 63 |
| 12.1 | Good Clinical Practice | 63 |
| 12.2 | Data Monitoring Committee | |
| 12.3 | Institutional Review Board/Independent Ethics Committee | 63 |
| <b>12.4</b> | Informed Consent | 63 |
| 12.5 | Records Management | 64 |
| 12.5.1 | Source Documentation | |
| 12.5.2 | Study Files and Record Retention | 64 |
| <b>12.6</b> | Conflicts of Interest | |
| | ATA MANAGEMENT, AUDITING, AND MONITORING | |
| 13.1 | Data Management | |
| 13.2 | Auditing | |
| 13.3 | Monitoring | |
| 14 A | MENDMENTS | 68 |
| | FUDY REPORT AND PUBLICATIONS | |
| | FUDY DISCONTINUATION | |
| | ONFIDENTIALITY | |
| | EFERENCES | |
| | PPENDICES | |
| 19.1 | APPENDIX I – Names of Study Personnel | |
| 19.2 | APPENDIX II – Adverse Event Intensity Grading | |
| 19.3 | APPENDIX III – Cytochrome P450 2B6, 2C8, 2C9, and 2D6 Substrates | 95 |
| | LIST OF TABLES | |
| Table | 1 Schedule of Assessments | 37 |
| Table | | |
| Table | | |
| <b>Table</b> | • | |
| | in HBV DNA levels at Week 12 or 24 between Treatment Groups | |
| | LIST OF FIGURES | |
| Figure | 21 Study Schematic | 36 |

#### LIST OF ABBREVIATIONS AND TERMS

AFP alpha fetoprotein

ALT alanine aminotransferase

API active pharmaceutical ingredient

AST aspartate aminotransferase

BMI body mass index

CC<sub>50</sub> 50% cytotoxic concentration cccDNA covalently closed circular DNA CFR Code of Federal Regulations CHB chronic hepatitis B infection

CI confidence interval

CKD-EPI Chronic Kidney Disease Epidemiology Collaboration

C<sub>max</sub> maximum plasma concentration

CNS central nervous system

CpAM core protein allosteric modifier

CRO Contract Research Organization (PRA Health Sciences)

CYP cytochrome P450
DAA direct acting antivirals
DAIDS Division of AIDS

DMC Data Monitoring Committee

dsDNA double-stranded DNA

EC<sub>50</sub> 50% effective concentration

ECG electrocardiogram

eCRF electronic case report form EDC electronic data capture

ETV entecavir

FSH follicle-stimulating hormone
GCP Good Clinical Practice
GFR glomerular filtration rate
GLP Good Laboratory Practices
GMP Good Manufacturing Practices

HAV hepatitis A virus HbA1c hemoglobin A1c

HBcAb antibody to the HBV core protein HBCrAg hepatitis B core-related antigen

HBeAb HBeAg antibody
HBeAg hepatitis B "e" antigen
HBsAb HBsAg antibody

HBsAg hepatitis B surface antigen

HBV hepatitis B virus

HCC hepatocellular carcinoma

HCV hepatitis C virus
HDV hepatitis D virus
HEV hepatitis E virus

HIV human immunodeficiency virus

IB Investigator's Brochure ICF Informed Consent Form

ICH International Council for Harmonisation

IEC Independent Ethics Committee

IFN interferon

IgM immunoglobulin M

INR International Normalized Ratio IRB Institutional Review Board

ISG IFN-stimulated gene

ITT intent-to-treat
IUD intrauterine device
LLN lower limit of normal
LOQ limit of quantitation

MedDRA Medical Dictionary for Regulatory Activities

MRI magnetic resonance imaging
NOAEL no-observed-adverse effect level

NUC nucleos(t)ide inhibitors of the HBV polymerase; also called nucleos(t)ide

analogues or nucleos(t)ides

PBMC peripheral blood mononuclear cell

pgRNA pre-genomic RNA PK pharmacokinetic(s)

PK1 Pharmacokinetic Population 1
PK2 Pharmacokinetic Population 2
Pol/RT polymerase/reverse transcriptase

PP per-protocol RBC red blood cell

rcDNA relaxed circular DNA SAP statistical analysis plan

SOC standard of care

Sponsor Assembly Biosciences

TDF tenofovir disoproxil fumarate

 $T_{max}$  time to  $C_{max}$ 

ULN upper limit of normal WHO World Health Organization

#### 2 INTRODUCTION AND RATIONALE

#### 2.1 Study Rationale

Worldwide >240 million people are chronically infected with the hepatitis B virus (HBV), and chronic hepatitis B infection (CHB) is a major global cause of severe liver morbidity and liver-related mortality [WHO, 2015]. Moreover, the burden of global mortality attributable to chronic viral hepatitis (B and C combined) has increased over the last two decades; it was the seventh leading cause of death worldwide in 2013, compared with the tenth in 1990 [Stanaway 2016]. Current therapies (comprising interferon [IFN] products and nucleos(t)ide inhibitors [NUCs] of the HBV polymerase) are highly effective at suppressing serum viremia but rarely lead to loss of viral antigenemia – a biomarker of persistent covalently closed circular DNA (cccDNA) activity. Additionally, in a surprising number of patients, ongoing low-level viremia remains detectable, as does cccDNA and intrahepatic viral intermediates [Boyd 2016; Marcellin 2014]. As a result of the persistence of active cccDNA, durable antiviral response is rare after cessation of treatment [Papatheodoris 2016]. New therapies are required which can increase functional cures, either alone or in combination with existing standard of care (SOC) for CHB.

ABI-H0731 is a novel HBV core protein allosteric modifier (CpAM) discovered by Assembly Biosciences ("the Sponsor"), and it is being developed as a potential therapeutic advance for CHB patients. ABI-H0731 inhibits HBV replication by interfering with essential functions of the HBV core protein, and it therefore inhibits HBV replication by different mechanisms than NUC analogues or IFN-α. In pre-clinical models, ABI-H0731 binds to the HBV core protein and induces altered, non-functional core protein assembly. Experience in patients with hepatitis C virus (HCV), another viral hepatitis, has shown that combination of multiple direct acting antivirals (DAAs) can increase rates of cures compared to monotherapy with a potent NUC inhibitor alone [Gane 2013]. Thus, inhibition of HBV core protein functions by ABI-H0731, when used in combination with currently approved HBV antivirals, may offer the potential to improve therapy for chronic HBV and provide patients with enhanced rates of functional cures in a finite treatment period.

This Phase 2a study will be the first study to explore the potential to increase rates of functional cure by addition of ABI-H0731 (a CpAM) to SOC NUC therapy, entecavir (ETV), in treatment-naïve, hepatitis B "e" antigen positive (HBeAg) positive CHB patients.

#### 2.2 Background

#### 2.2.1 Chronic Hepatitis B Virus

HBV remains a major public health burden. HBV contributes to as much as 30% of cases of cirrhosis and 45% of cases of hepatocellular carcinoma (HCC) [WHO 2015]. The standard serologic markers of HBV infection include: HBV DNA, HBsAg, antibody to HBsAg (HBsAb), HBeAg, antibody to HBeAg (HBeAb), and, in almost all patients, antibody to the HBV core protein (HBcAb). Chronic HBV infection is clinically defined as the persistence of HBsAg in a subject for 6 to 12 months or more [Heimbach 2018].

There are four major HBV genotypes (A, B, C, and D). Genotype A is regarded as pandemic and is predominantly found in North America, Northern/Western Europe, and Central Africa. HBV genotype

B is most common in Asia including China, Vietnam, Japan, Taiwan, and Indonesia. Genotype C is predominant in East Asia and Oceania. Genotype D (also pandemic) is most highly prevalent in North America, Asia (including India), the Mediterranean, India, and the Middle East [Guettouche and Hnatyszyn, 2005].

Despite broad implementation of HBV vaccination programs, new cases of HBV infection are still common. The World Health Organization (WHO) estimates that there are >4 million acute HBV infections worldwide each year [WHO 2015]. The global prevalence of chronic HBV infection shows wide geographic variation, with a prevalence of >8% people in highly endemic regions (eg, East Asia and equatorial Africa), 2% to 7% people in moderately endemic regions (eg, the Middle East and the Indian subcontinent), and <2% in locales of low endemicity (eg, North America and Europe) [WHO 2015].

Some HBV carriers will lose detectable serum HBsAg and HBV viremia will drop to non-detectable levels. Such a transition to an HBsAg-negative, minimally replicative state (termed "HBsAg seroconversion") is usually durable and, if it precedes the development of cirrhosis and HCC, is associated with improved long-term clinical outcomes [EASL 2012]. As such, HBsAg seroconversion is considered a "functional cure" and a potential endpoint for HBV therapy.

Currently there are two clinically accepted options for the treatment of CHB: IFNs and oral NUCs, which act as inhibitors of the viral polymerase. Of these, oral NUCs are much more broadly used, and have shown remarkable success in achieving maintained viral suppression in CHB patients, with associated decreases in long-term clinical complications [Liaw 2012]. Despite suppression of viremia for extended periods of time, however, HBsAg loss and/or seroconversion is rarely achieved in a practical timeframe with current therapies. HBsAg loss is achieved by <10% of CHB patients within 5 years after a year of treatment with IFN products and/or after 5 years of NUC antivirals, with slightly higher rates of HBsAg loss recently reported in combination studies of tenofovir disoproxil fumarate (TDF) together with pegylated IFN-alfa for one year [Marcellin 2014].

There is clearly a need for improved HBV therapies that are of finite duration and can produce a substantially higher rate of therapeutic responses that will be durable post-treatment. Specifically, improved rates of two types of durable outcomes are desirable for new HBV therapies: durable HBeAg loss/seroconversion (in HBeAg-positive patients), and HBsAg loss/seroconversion (in all patients), in addition to sustained off-treatment viral load suppression and normalization of transaminases. Such 'functional cures' are predicted to afford improved long-term patient outcomes, ie, reduced HBV-associated morbidity and mortality from end-stage liver disease and HCC.

## 2.2.2 Hepatitis B Virus Biology and Rationale for Hepatitis B Virus Core Protein Allosteric Modifiers (CpAMs)

#### 2.2.2.1 Overview of Hepatitis B Virus Biology

HBV is a member of the *Hepadnaviridae* family. The HBV genome consists of a partially double-stranded DNA (dsDNA) (~3.2 kb) that is synthesized through reverse transcription of its pre-genomic RNA (pgRNA) precursor. The infectious HBV virion, called the Dane particle, comprises an enveloped nucleocapsid, which contains a single copy of the HBV genome as partially double-stranded, relaxed

circular DNA (rcDNA) and viral reverse transcriptase, enclosed in a polymeric capsid, assembled from HBV core protein subunits. The life cycle of HBV can be conceptualized as occurring in several steps. Circulating HBV must enter cells. Following entry, virus must enter the nucleus where rcDNA is converted to a stable chromosome-like moiety (the cccDNA). The cccDNA functions as the template for full length pgRNA and the mRNAs for viral proteins. These proteins include polymerase/reverse transcriptase (Pol/RT), HBV X protein, core protein, and HBsAg. RNA produced from the cccDNA is transported from the nucleus into the hepatocyte cytoplasm, where it is bound by HBV polymerase and encapsidated by 120 viral core protein dimers. Within the capsid, pgRNA is reverse transcribed into viral dsDNA. This dsDNA filled particle can then either acquire an S antigen envelope and be secreted as new infectious virus or recycle rcDNA back to the nucleus where it can amplify the cccDNA pool. Details of the HBV replication cycle have recently been reviewed in detail by Seeger et al [Seeger 2013].

#### 2.2.2.2 Hepatitis B Virus Core (Capsid) Protein and Core Protein Functions

HBV core protein has several essential roles in the life cycle of HBV infection, including the formation of capsids. The appropriate kinetics of HBV core protein assembly is critical in enabling functional capsid formation and encapsidation of pgRNA. These steps are essential for the formation of new infectious virions. The HBV capsid is also essential for the process of nuclear import of the HBV rcDNA through a regulated interaction with nuclear pore proteins. In the nucleus, the rcDNA is converted to cccDNA. cccDNA is a long-lived circular, episomal DNA from which all HBV RNAs are derived. Core protein contributes to replenishing nuclear cccDNA pools by mediating nuclear import of genomic DNA from newly formed capsids in the cytoplasm of infected cells. Nuclear forms of HBV core protein can also affect the expression of viral and host genes and contribute to regulated splicing and nuclear export of HBV RNAs, and HBV CpAMs have been reported to be able to interfere with cccDNA function [Gruffaz 2013, Belloni 2013]. HBV core protein is therefore a critical component of the HBV life cycle. Additionally, some data suggest that HBV core protein induces an HBV-specific dysfunction of the innate immune response in HBV-infected hepatocytes [Gruffaz 2013], including a suppression of expression of IFN-stimulated genes (ISGs).

These findings suggest that allosteric modulation of core protein may allow targeting of multiple aspects of the viral life cycle: assembly into virion capsids, trafficking of HBV DNA into cell nuclei, cccDNA replenishment, and potentially interference with the innate immune response in infected cells.

#### 2.2.2.3 Hepatitis B Virus Core Protein Allosteric Modifiers and ABI-H0731

#### 2.2.2.3.1 *In Vitro* Activity of ABI-H0731

ABI-H0731 is a small molecule inhibitor of HBV replication that induces non-functional assembly of the HBV core protein and exhibits potent inhibition of HBV replication *in vitro* via a different mechanism than NUC or IFN- $\alpha$  therapy. ABI-H0731 binds to the HBV core protein and induces altered, non-functional core protein assembly *in vitro*. The antiviral activity of ABI-H0731 against HBV replication *in vitro* was evaluated using a standard HepAD38 cell line, which stably expresses infectious genotype D HBV. Analysis of intracellular HBV DNA showed a dose-dependent reduction of viral DNA in the presence of ABI-H0731. In an inducible cell line model of HBV, the mean 50% effective concentration (EC<sub>50</sub>) for ABI-H0731 against HBV DNA replication was 173 nM, with no cellular toxicity observed at the highest concentration tested (50% cytotoxic concentration [CC<sub>50</sub>] >10  $\mu$ M).

Similar or better antiviral activity (EC<sub>50</sub> of 86-142 nM) was observed in HBV DNA transfection-based assays against representative HBV strains of genotypes A, B, C, and D. ABI-H0731 therefore showed broad inhibition across genotypes.

Specificity of ABI-H0731 for HBV was confirmed by the absence of antiviral activity when tested against other DNA and RNA viruses (HSV-1, HRV-16, and influenza A) at the highest concentrations tested (10  $\mu$ M). ABI-H0731 was also evaluated for selectivity by determining the CC<sub>50</sub> levels in seven human cell types/lines (Huh7, HepG2, HeLa H1A, HEK 293, NCI H226, and MOLT-4) and freshly isolated peripheral blood mononuclear cell (PBMC) cultures representing various human tissues following 4 days of incubation. ABI-H0731 showed no significant effects at a concentration of 3.3  $\mu$ M (<7% reduction in cell viability) and up to 16% reduction in cell viability in some cell types/lines at 10  $\mu$ M. These results demonstrate that ABI-H0731 is a highly selective and specific HBV inhibitor, consistent with specificity in targeting the HBV core protein target of ABI-H0731.

See the Investigator's Brochure (IB) for further information.

#### 2.2.2.3.2 <u>Combination Therapy</u>

Combining drugs from different classes provides numerous advantages compared with monotherapy, including the potential for additive or synergistic antiviral effects and establishment of higher resistance barriers, reducing the likelihood of adverse mutations. Combination studies of ABI-H0731 with a representative NUC polymerase inhibitor, ETV (Baraclude®), showed additive to synergistic effects over a wide range of concentrations, with no evidence of antagonism, indicating that ABI-H0731 has the capacity to be successfully combined with NUCs in the treatment of HBV. Please see the IB for further information.

#### 2.2.2.3.3 Study Drug Resistance

There are no established methods for the selection of drug resistance against HBV *in vitro* because there are no *in vitro* cell culture systems that allow multiple cycles of HBV replication. In the Phase 1b monotherapy study, ABI-H0731-101(b), CHB subjects treated with ABI-H0731 for 28 days were monitored closely for evidence of resistance emergence. To date, a single subject was observed to enter study ABI-H0731-101(b) harboring a resistance variant at baseline (T109M). While this subject had a blunted response to therapy, they still exhibited a 1 log<sub>10</sub> IU/mL decline in viral load over 28 days, suggesting that ABI-H0731 may achieve sufficient intrahepatic concentrations to inhibit replication of at least some naturally occurring resistant mutants. Importantly, the T109M mutant is not known to have a reduced susceptibility to SOC NUCs or pre-exist as a polymorphic substitution in HBV database sequences at any significant frequency. To date, no *de novo* mutations were noted to arise on treatment in any other subjects.

#### 2.2.3 Summary of Nonclinical Pharmacology and Toxicology

The nonclinical pharmacokinetics (PK), absorption, distribution, metabolism, and excretion of ABI-H0731 were characterized *in vitro* and *in vivo* in mice, rats, dogs, rabbits, and monkeys. Results are summarized in the IB.

A standard battery of nonclinical safety studies, including safety pharmacology, genotoxicity, and *repeat* dose toxicity studies has been conducted. In safety pharmacology studies, there were no adverse central nervous system (CNS), cardiovascular, or respiratory system effects in rats or monkeys following single oral doses of ABI-H0731 up to 500 mg/kg. ABI-H0731 was not genotoxic in the *in vitro* bacterial or mammalian cell assays or in the *in vivo* rat micronucleus study.

In chronic toxicity studies, ABI-H0731 was well-tolerated at the highest tested dose levels of 250 mg/kg/day for 6 months in rats and 500 mg/kg/day for 9 months in monkeys, with no drug-attributed animal deaths and no patterns of adverse effects or changes in clinical pathology. There were no clear target organ findings in these studies. Histopathology observations in rats consisted of increased adrenal gland weight for males given  $\geq 100$  mg/kg/day and females given  $\geq 200$  mg/kg/day, with correlating microscopic findings of minimal or mild diffuse hypertrophy of the zona fasciculata and/or minimal to moderate multifocal cortical vacuolation in some animals given  $\geq 100$  mg/kg/day. These findings were considered non-adverse, based on the absence of any apparent detrimental effect on the overall health of the animals and the partial or complete reversibility of the effects during the 28-day recovery period. In monkeys, there were no measurable effects beyond normal morphologic variations. Therefore, the no-observed-adverse effect levels (NOAELs) are the highest doses tested, 250 mg/kg/day for 6 months in rats and 500 mg/kg/day for 9 months in monkeys. These dosing levels resulted in rat and monkey maximum plasma concentrations ( $C_{max}$ ) levels of 10.0 µg/mL and 8.47 µg/mL, respectively, and area under the concentration-time curve from time 0 to 24 hours post-dose values of 147 hr\*µg/mL and 122 hr\*µg/mL, respectively. For more information, please refer to the IB.

#### 2.2.4 Summary of Clinical Studies with ABI-H0731

Clinical Experience with ABI-H0731 consists primarily of three early-phase clinical studies: (1) the recently completed Phase 1a/1b dose-ranging study in healthy volunteers and treatment-naïve CHB subjects, ABI-H0731-101; (2) an essentially identical sister Phase 1b study ABI-H0731-101B (in treatment-naïve subjects with CHB); and (3) the second recently completed Phase 1a study ABI-H0731-102. These studies are summarized briefly below. For more complete information, please refer to the IB.

#### 2.2.4.1 Clinical Safety Data of ABI-H0731

Clinical experience with ABI-H0731 consists of two Phase 1 dose-ranging studies conducted to assess the safety, tolerability, PK, and initial efficacy of ABI-H0731 monotherapy:

- The first-in-human study Phase 1a conducted in healthy volunteers in New Zealand (ABI-H0731-101, Part 1). Intensive PK was assessed following single ascending doses (100, 300, 600, and 1,000 mg) under fasted (100 and 300 mg) and fed (300, 600, and 1,000 mg) conditions, as well as 800 mg once daily and 800 mg twice daily (under fed conditions) for 7 days. Overall, the results suggested that these single and multiple oral doses of ABI-H0731 were well-tolerated with dose-related increases in plasma exposures. During the off-treatment follow-up period, one subject in the 800 mg once daily cohort and two subjects in the 800 mg twice daily cohort developed transient rashes that were considered mild (Grade 1).
- A Phase 1b study conducted at multiple sites in Australia, New Zealand, Hong Kong, England, South Korea, and Taiwan (ABI-H0731-101, Part 2, and ABI-H0731-101B) in which HBV patients received

ABI-H0731 at doses of 100, 200, 300, or 400 mg once daily for 28 days. ABI-H0731 was well-tolerated in CHB subjects at 100, 200 and 300 mg once daily through the 28-day dosing period and two weeks of follow-up (follow-up out to 4 weeks post-treatment is ongoing at the time of this IB update). One subject in the 300 mg cohort developed a transient localized (Grade 1) rash approximately two days following the end of therapy. The rash was considered unrelated to drug both by the Investigator and a consulting dermatologist. One of two subjects dosed in the 400 mg once daily cohort developed a Grade 3 rash following 10 days of dosing. The rash was deemed related to study drug, and the subject was discontinued from treatment. The rash rapidly resolved off treatment with no other intervention required. Other than the individual subject with the Grade 3 rash, all other treatment-emergent adverse events were considered mild (Grade 1), and all Phase 1b subjects completed their study dosing and follow-up evaluations. There were no other premature treatment-emergent laboratory abnormalities that were deemed drug related and clinically significant.

• A Phase 1a study conducted in healthy volunteers in the US to obtain additional safety and PK data for a longer dosing period (ABI-H0731-102). Three cohorts received ABI-H0731 at 100 mg, 200 mg or 300 mg once daily for 14 days. Treatment-emergent adverse events were infrequent (six in total), mild, and deemed unrelated to study drug. Laboratory abnormalities were generally minor, not related to dose, duration or target organ, and considered not clinically significant. PK data were consistent with the previous Phase 1a study.

For more complete information, please refer to the IB.

#### 2.2.4.2 Preliminary Pharmacokinetic Data for ABI-H0731

PK parameters from studies ABI-H0731-101 and ABI-H0731-102 were calculated from plasma concentration over time, using WinNonlin<sup>TM</sup> software. In general, ABI-H0731 was rapidly and well absorbed following oral administration, with a median time to maximum plasma concentration (T<sub>max</sub>) ranging from 3 to 4.5 hours. ABI-H0731 demonstrated increasing exposures as doses increased, which were approximately dose proportional with modest variability through 600 mg, and it exhibited a terminal half-life of approximately 24 hours. Clinical activity was seen with the lowest doses explored (100 mg).

Based on the pre-dose trough assessments in ABI-H0731-101, ABI-H0731-101(b), and ABI-H0731-102 protocols, it appears that PK steady-state may be achieved by or prior to Day 5. Detailed information can be found in the IB.

#### 2.3 Risk/Benefit Assessment

#### 2.3.1 Known and Potential Risks of ABI-H0731

ABI-H0731 is a novel direct acting HBV inhibitor that will be among the first HBV CpAMs to be investigated in CHB subjects for > 28 days. At this stage of development, the risk considerations for ABI-H0731 are primarily based on the non-clinical and Phase 1 data summarized in the IB.

No evidence was found for genotoxicity or clastogenicity.

In the Good Laboratory Practices (GLP) chronic toxicology studies in rats and monkeys, ABI-H0731 was generally well-tolerated, with no animal deaths or severe in-life effects attributed to ABI-H0731 treatment at any exposure level (refer to the IB). There were no clear target organ findings in these studies, and the NOAELs were the highest doses tested, 250 mg/kg/day for 6 months in rats and 500 mg/kg/day for 9 months in monkeys. Specialized safety pharmacology studies were conducted to the same maximal dosing intensities as the 28-day GLP toxicology studies, 500 mg/kg/day in rats and 300 mg/kg/day in monkeys, with the results indicating no appreciable adverse effects on cardiac, respiratory, or CNS functions at any ABI-H0731 dose level.

Human exposure data for ABI-H0731 was obtained from the three Phase 1 clinical studies described above, in which a total of 84 healthy volunteers, and 38 CHB subjects were treated with ABI-H0731 or matching placebo (refer to the IB). The single- and multiple-dose exposures were closely monitored with clinical and laboratory assessments at each study visit. ABI-H0731 was well-tolerated with no serious adverse events, no clinically significant vital sign or electrocardiogram (ECG) changes, and no treatment-emergent drug related clinically significant laboratory findings. One CHB subject was discontinued from treatment because of a Grade 3 rash, which resolved with no further intervention required other than drug discontinuation. Across all studies, with the possible exception of rash, there was no pattern of adverse events nor of laboratory abnormalities that suggested any potential target organ pathology was associated with either dose or duration of ABI H0731 exposure.

Refer to the IB for additional information.

#### 2.3.2 Known and Potential Benefits of ABI-H0731

There is a need for improved HBV antiviral therapies that can offer a "functional cure" for patients with CHB. Such therapy should produce durable post-treatment suppression of viral load and normalization of transaminases, and, ideally, a loss of detectable viral antigens in a higher proportion of CHB patients than achieved with current therapies. The HBV core protein is involved in multiple aspects of the HBV life cycle. Therapy with CpAMs may disrupt multiple core protein functions (including cccDNA replenishment and possibly core-mediated interactions with HBV-specific immune responses) and thus is a highly attractive class of novel DAAs that may increase functional cure rates for CHB.

In Phase 1a and 1b studies, ABI-H0731 has been able to safely achieve liver and blood levels sufficient to demonstrate significant antiviral activity. The resultant decrease in detectable HBV DNA and RNA in serum or plasma supports inhibition of RNA packaging and is consistent with the mechanism of action – inappropriate polymerization of HBV core protein. It is anticipated that this pleotropic mechanism of action may lead to more complete inhibition of the viral replicative cycle than inhibition of the viral polymerase alone, resulting in more rapid loss of active cccDNA and higher rates of functional cures for CHB patients.

This study will specifically evaluate a 6-month course of therapy that may provide a lasting therapeutic benefit. Subjects who complete this study will be offered the opportunity to enroll into an open-label, extension study of ABI-H0731 treatment with SOC NUC therapy. In the extension study, all subjects will receive up to 12 additional months of ABI-H0731.

#### 2.3.3 Assessment of Potential Risks and Benefits

In this study, chronically HBV-infected adults who have not previously been treated for HBV >4 weeks with a NUC or with any CpAM other than ABI-H0731 will be enrolled. These subjects will have detectable viremia as well as circulating biomarkers of ongoing viral replication and active cccDNA transcription – HBsAg, HBeAg, hepatitis B core-related antigen (HBCrAg), and encapsidated viral RNA. The 24-week treatment period in this Phase 2a trial is expected to be sufficient to assess the safety and tolerability of ABI-H0731 + ETV combination therapy as well as the potential for increased rate of functional cure via more rapid reduction in viral load and increased loss of active cccDNA as compared to subjects on ETV therapy alone.

As compared to monotherapy with ETV alone, addition of ABI-H0731 is expected to result in more complete suppression of cccDNA metabolism and pleotropic effects on the viral core protein, potentially resulting in accelerated loss of cccDNA. ABI-H0731 with ETV therapy is thus anticipated to demonstrate clinical antiviral effects not seen with ETV monotherapy (eg, serum HBV RNA, HBsAg, and HBeAg reductions). The degree of reduction or duration of effect with 24 weeks of therapy, however, may be insufficient to establish any lasting clinical benefit for any of the subjects enrolled. The predictable benefits of this study are thus primarily the clinical care provided as a part of this clinical study, the potential benefit derived from the ETV therapy provided as part of this study, as well as the potential for additional benefit if ABI-H031 with ETV therapy does increase rates of cccDNA loss.

Eligible subjects will also be provided the opportunity to enroll into a long-term, open-label, extension study (ABI-H0731-211) to evaluate if longer courses of combination therapy (with ETV and ABI-H0731) increase the potential for functional cure. Subjects who choose not to enroll in the long-term extension study will continue to be followed for up to 12 more weeks on ETV alone as part of this study (ABI-H0731-202). After the 12-week follow-up period, subjects may elect to continue on ETV or other SOC therapy in consultation with their Study Investigator or external treating physician. Subjects who choose not to continue on SOC therapy after completion of 3-month follow-up should be monitored closely for the potential for viral rebound and possible "flare" with associated decompensation. Risk of such a flare is mitigated by the recommendation for SOC therapy and careful patient selection for inclusion into this protocol. Additionally, any follow-on treatment required for management of a post-treatment ALT flare, as defined in this protocol, will be reimbursable by the Sponsor for up to one-year post-study.

#### 3 STUDY OBJECTIVES AND ENDPOINTS

#### 3.1 Objectives

#### 3.1.1 Primary Objective

To evaluate the potential for ABI-H0731 to increase the rapidity of HBV DNA loss in HBeAgpositive CHB subjects by initiating treatment with ABI-H0731 + ETV in subjects who are not yet on treatment for CHB, as measured by timing and magnitude of change in serum HBV DNA from Baseline

#### 3.1.2 Secondary Objectives

- To evaluate the safety and tolerability of ABI-H0731 in combination with ETV therapy as initial therapy for HBeAg-positive CHB subjects
- To confirm a lack of drug-drug interactions between ETV and ABI-H0731
- To evaluate the potential for emergence of resistance, if any, for ABI-H0731 in combination with ETV therapy

#### 3.1.3 Exploratory Objectives

- To evaluate the kinetics of and absolute changes from Baseline in biomarkers of transcriptionally active cccDNA (HBeAg and HBsAg)
- To evaluate the kinetics of and absolute changes from Baseline in circulating viral RNA
- To assess the relationship between exploratory viral biomarkers such as changes in viral RNA and HBCrAg and outcome
- To explore the PK of ABI-H0731
- For subjects who provide an optional pharmacogenomic sample, to evaluate the potential contribution of host genomics to outcomes

#### 3.2 Study Endpoints

#### 3.2.1 Primary Endpoint

The primary efficacy endpoint will be:

• Change in mean  $log_{10}$  HBV DNA from Baseline (Day 1) to Week 12 or Week 24 on ABI-H0731 + ETV as compared to placebo + ETV

#### 3.2.2 Secondary Endpoints

Secondary endpoints will be:

- Number of subjects with adverse events, premature discontinuations, abnormal safety laboratory results, ECG, or vital signs
- Subjects with abnormal alanine aminotransferase (ALT) at Baseline who have normal ALT at Week 24 on ABI-H0731 + ETV as compared to placebo + ETV
- Percent of subjects with a decline in viral DNA to below limit of quantitation (LOQ; on ABI-H0731 + ETV as compared to placebo + ETV) at end of treatment
- Median time to viral suppression, defined as HBV DNA <20 IU/mL, on ABI-H0731 + ETV as compared to placebo + ETV
- Emergence of resistant HBV variants, if any
- Drug concentrations:
  - o Trough levels and (in subjects where optional samples are available) trough to peak ratios of ABI-H0731 on ABI-H0731 + ETV
  - o Trough levels and (in subjects where optional samples are available) trough to peak ratios of ETV on ABI-H0731 + ETV therapy as compared with placebo + ETV

#### 3.2.3 Exploratory Endpoints

Exploratory endpoints will include:

- Quantitative changes in serum viral antigen (HBsAg or HBeAg, and HBCrAg) on ABI-H0731 + ETV as compared with placebo + ETV, at each time point
- Subjects with loss (defined as below LOQ) or decline in HBsAg and or HBeAg (<0.5 log<sub>10</sub>, ≥0.5 to 1.0 log<sub>10</sub>, or >1.0 log<sub>10</sub> decrease in viral antigen) on ABI-H0731 + ETV as compared with placebo + ETV at end of treatment and end of follow-up
- Subjects with HBsAg or HBeAg seroconversion (loss of HBsAg and appearance of HBs antibody) or HBeAg seroconversion (loss of HBeAg and appearance of HBe antibody) on ABI-H0731 + ETV as compared with placebo + ETV
- Quantitative changes from Baselines in mean log<sub>10</sub> viral RNA, on ABI-H0731 + ETV, as compared with placebo + ETV, at each time point
- Subjects whose HBV DNA achieves "target not detected" on ABI-H0731 + ETV as compared with placebo + ETV

- For subjects who do NOT rollover onto the optional extension study ABI-H0731-211:
  - Subjects with suppression of detectable serum HBV RNA on treatment whose RNA rebounds after discontinuing investigational treatment with ABI-H0731 + ETV as compared with placebo + ETV therapy
  - Subjects with changes in HBsAg or HBeAg whose viral antigen rebounds off therapy after discontinuing investigational treatment with ABI-H0731 + ETV as compared with placebo + ETV therapy
  - Subjects with HBsAg or HBeAg loss at Week 24 that is maintained through end of follow-up (Week 36) after discontinuing investigational treatment with ABI-H0731 + ETV therapy as compared with placebo + ETV therapy
- If differences are seen in outcomes/adverse events between racial or ethnic groups: Pharmacogenomics correlation with clinical outcomes subjects who provide optional informed consent

#### 4 STUDY PLAN

#### 4.1 Study Design

This Phase 2a, multi-center, randomized, double-blind, placebo-controlled study will assess the safety, efficacy, PK, and pharmacodynamics of 300 mg ABI-H0731 daily in combination with ETV in treatment-naïve subjects with HBeAg-positive CHB. Subjects will be randomized 1:1 to receive investigational agent (ABI-H0731 + ETV or matching placebo + ETV) for up to 6 months. ETV will continue uninterrupted for the duration of the study as well as during follow-up.

Safety will be monitored by a Data Monitoring Committee (DMC), including a safety analysis after all subjects have completed Week 12 (or discontinued study without completing Week 12). There will be an assessment of PK data after all subjects have completed Week 4 (or discontinued study without completing Week 4) to confirm a lack of an important impact of ABI-H0731 on the steady-state PK of ETV.

At the end of the treatment period in this study, subjects will either continue ETV and stop treatment with ABI-H0731/placebo or they may elect to roll over onto the optional, open-label, extension study ABI-H0731-211.

- Subjects who do <u>not</u> roll over into the optional, open-label, extension study ABI-H0731-211 will be treated under the direction of their Study Investigator and monitored for an additional 12 weeks to determine if any changes in either viral antigens or viral RNA which may have been noted on treatment will persist through end of follow-up. Refer to Section 2.3.3 of this protocol for additional post-study follow-on guidance.
- Subjects who do elect to roll over to the optional, open-label, extension study of ABI-H0731 + SOC NUC (protocol ABI-H0731-211) will continue on open-label combination therapy as per that study. The objective of the study ABI-H0731-211 will be to evaluate the safety and potential for benefits of up to one additional year of therapy with ABI-H0731 in combination with SOC NUC therapy. Subjects will be required to sign a separate consent prior to entering the ABI-H0731-211 study.

#### 4.2 Scientific Rationale

It is anticipated that addition of ABI-H0731, a DAA targeting the HBV core protein to ETV, a SOC NUC therapy, will be safe and may result in an increase in the functional cure rate for subjects with CHB by preventing the establishment and possible maintenance of cccDNA more completely than ETV therapy alone. Combination therapy with two potent DAAs is expected to result in a more rapid decrease of viral DNA as compared to monotherapy, as well as a decrease of serum viral RNA. Additionally, combination therapy is expected to result in a greater loss of cccDNA with a corresponding decline in serum viral antigens which reflect the presence and activity of cccDNA (eg, HBsAg and HBeAg). This study will explore both the safety of combination therapy in HBeAg-positive, treatment-naïve subjects, as well as evaluate measures of antiviral efficacy such as reduction in serum viral DNA, reduction in circulating viral RNA, and potential serum biomarkers of functional cures: quantitative and qualitative reduction in the viral antigens HBeAg and HBsAg.

#### 4.3 Dose Justification

In the Phase 1 clinical studies, ABI-H0731 was well-tolerated in healthy subjects at daily doses up to 1000 mg, twice daily doses of 800 mg for 7 days, and at daily doses up to 300 mg for 14 days. All treatment-emergent adverse events were considered mild (Grade 1) and reversible. Similarly, in subjects with CHB, at doses up to 300 mg daily for 28 days, ABI-H0731 was well-tolerated and all drug related treatment-emergent adverse events were mild (Grade 1) and reversible. One subject with CHB developed a Grade 3 rash after approximately 10 days of repeated doses of 400 mg daily, the rash resolved off treatment with no intervention required other than dose discontinuation.

Preliminary data indicated that there is a dose-dependent decrease in viral load at doses of 100 mg, 200 mg, and 300 mg daily in subjects with CHB. It is expected that 300 mg daily will be safe and provide sufficient exposure to ABI-H0731 to produce the desired antiviral effect i within the dose range that was well-tolerated in healthy subjects and subjects with CHB.

#### 4.4 Study Drug Resistance Monitoring

To assess potential HBV core gene sequences associated with viral resistance or blunted treatment response, serum samples from subjects with evidence of nonresponse to treatment, viral DNA rebound (>1  $\log_{10}$  HBV DNA rebound from on treatment nadir) or viral load plateauing ( $\geq 2$  consecutive samples with viral load remaining within 0.5  $\log_{10}$  of nadir) will be selected for HBV core gene sequencing, with sequence comparisons to baseline sequences, as well as comparisons to core gene sequences from placebo recipients and HBV database sequences.

#### 4.5 End of Study Definition

The study will be completed when the last subject completes the 12-week, post-treatment follow-up period, or when the last subject transitions to protocol ABI-H0731-211, or when the last subject discontinues study before completing the follow-up period or transitioning to the extension study, whichever is later.

#### 4.6 Management of Toxicities

#### 4.6.1 Subjects with Alanine Aminotransferase Elevations

Subjects experiencing ALT elevations  $\geq$  2×Baseline or on-treatment nadir and >2×upper limit of normal (ULN) during study treatment or during post-treatment follow-up will be closely monitored. The following guidance is offered for management of study subjects with ALT elevations or biochemical evidence of declining hepatic function:

#### • ALT flare on treatment

o All subjects with an ALT flare on treatment, defined as ALT > 2×Baseline or on-treatment nadir and ≥10×ULN, should have the ALT findings confirmed within 3 days of receipt of the original results. All subjects should return for an unscheduled visit and undergo a symptom directed physical examination, review of concomitant medications (including herbal medications or

supplements), and the following laboratory tests: ALT, aspartate aminotransferase (AST), total bilirubin, International Normalized Ratio (INR), and serum albumin. If the ALT flare is confirmed, HBV DNA, quantitative HBV serologies (HBeAg [reflex qualitative HBeAg if quantitative HBeAg is negative] and HBsAg [reflex qualitative HBsAg if quantitative HBsAg is negative]), hepatitis A virus (HAV) immunoglobulin M (IgM), HCV RNA, hepatitis D virus (HDV) RNA, and hepatitis E virus (HEV) IgM should also be drawn.

- If an intercurrent cause is determined to be causal, the intercurrent cause should be treated as deemed medically appropriate by the treating physician.
- In the absence of evidence of declining hepatic function, and in the absence of contraindications, subjects with an ALT flare may continue on study under close observation.
  - o If ALT is rising at the confirmatory visit, subjects should return for an unscheduled visit every 2-5 days until the ALT elevation has stabilized. Subjects whose ALT has stabilized should continue to be monitored weekly (or more frequently as deemed necessary by the treating physician) until ALT values return to normal or baseline levels.
- Subjects with ALT "flares" or ALT elevations without declining hepatic function or contraindications should stop study drug if the ALT remains persistently elevated for > two weeks in the absence of decreasing HBV DNA (if detectable), and/or HBV RNA, and/or viral antigen (HBeAg or HBsAg).
- Declining hepatic function during treatment
  - O Subjects with confirmed biochemical evidence of declining hepatic function, should be discontinued from study treatment. Declining hepatic function is defined as:
    - ALT elevation  $\ge 2 \times \text{Baseline}$  or nadir and  $\ge 2 \times \text{ULN AND}$ 
      - o Direct bilirubin increase to  $\ge 2 \times \text{Baseline}$  and  $\ge 2 \times \text{ULN OR}$
      - An albumin decline  $\ge 0.5$  g/dL OR INR  $\ge 2 \times$ Baseline OR
      - Symptoms of liver inflammation (fatigue, weakness, lack of appetite, nausea, vomiting, jaundice or discolored feces)
  - O Subjects with evidence of declining hepatic function should return for an unscheduled visit every 2-5 days until the relevant laboratory values stabilize. Subjects whose hepatic function has stabilized should continue to be monitored weekly (or more frequently as deemed necessary by the treating physician) until the relevant laboratory values return to normal or baseline.
- Post-treatment ALT "flare" or ALT elevation with declining hepatic function
  - o For subjects who elect not to enroll in the open-label extension study ABI-H0731-211, risk of post-treatment flare is mitigated by advising subject to continue on ETV for their CHB. Any

subject with a post-treatment ALT elevation meeting the ALT "flare" definition or a lesser post-treatment ALT elevation with biochemical evidence of declining hepatic function (described above), while on treatment with a regulatory-approved HBV antiviral agent should return for an unscheduled visit every 2-5 days until the relevant laboratory values stabilize. Subjects whose hepatic function has stabilized should continue to be monitored weekly (or more frequently as deemed necessary by the treating physician) until the relevant laboratory values return to normal or baseline. Subsequently, subjects should continue to be followed on their regular study visit schedule, with the addition of any unscheduled visits the Principal Investigator believes are merited for the safety and well-being of the subject.

All subjects with declining hepatic function or ALT flare (on or off treatment) should continue to be followed on their regular study visit schedule, with the addition of unscheduled visits as described above. If the post-treatment ALT flare has not substantially resolved by the last study follow-up visit, subjects should continue to return to clinic as deemed medically appropriate by the Principal Investigator, in consultation with the Sponsor, and the unscheduled visit module in the case report form should be utilized as needed to gather additional clinical and laboratory data until the ALT flare is documented to be either resolved or resolving (defined as consistent ALT declines of 10% or more or normalization of ALT) on at least two successive visits.

If 2 or more subjects meet these LFT flare management criteria, the US FDA and other relevant regulatory agencies will be notified.

#### 4.6.2 Subjects with Rash

In the event of any rash, subjects should return to clinic for evaluation for an unscheduled visit (Day 0 of rash). Digital photographs of the rash should be taken, and blood samples should be taken and evaluated at the site's local laboratory as well as the central laboratory. Laboratory tests should include: erythrocyte sedimentation rate, complete blood count (with differential), creatinine, ALT, AST, and total bilirubin. Local laboratory reports and digital photographs will be de-identified, collected by the site monitor, and securely stored by the Sponsor.

If the rash diagnosis is uncertain, or if a rash is Grade 2, a referral to a dermatologist should be made and a skin biopsy should be conducted if recommended by the dermatologist. For a rash that is Grade 3 or higher, a referral to a dermatologist should be made and a skin biopsy should be requested of the dermatologist. All dermatologist reports and skin biopsy results will be included in the source and electronic case report form (eCRF). A copy of the dermatologist report will be de-identified and collected by the monitor on behalf of the Sponsor.

If the rash is considered by the Investigator to be likely related to a non-study exposure (drug, food, or concomitant illness), then subjects should be treated symptomatically and as deemed appropriate by the Investigator (or consulting dermatologist) until the rash has resolved. Additional unscheduled visits should be performed during the study at the Investigator's prerogative until resolution of the rash. Digital photographs of lesions should be obtained at each visit to document any change in condition. If required for subject management, local and central laboratory samples should also be drawn at additional unscheduled visits. Any local laboratory test results and digital photographs will be de-identified,
collected by the site monitor, and securely provided to PRA Health Sciences ("the Clinical Research Organization [CRO]") for provision to the Sponsor.

If rash is considered possibly or probably related to study drug, then:

- For Grade 1 rashes, subjects can continue to take study drug at the Investigator's discretion
- For Grade 2 rashes, subjects may continue to take study drug in consultation with Sponsor and at the Investigator's discretion. If the rash progresses or worsens, subjects must discontinue study drug. Subjects should be advised to contact the study site staff immediately if the rash worsens, if systemic signs develop, or if mucosal lesions develop
- For Grade 3 and higher rashes, study drug will be discontinued and the subjects will continue on study as described below

Subjects with rashes should continue to be followed on their study visit schedule even if treatment is discontinued, with additional unscheduled visits as deemed medically appropriate by the Investigator.

If the rash has not substantially resolved by the last study visit, subjects should return for an unscheduled visit at least every other week or as deemed medically appropriate by the Investigator. Unscheduled visits should continue until the rash has resolved or declined to Grade 1 or less for two successive visits.

## 4.7 Study Schematic

The study schematic is presented in Figure 1.

Figure 1 Study Schematic



I/E = inclusion/exclusion

#### 4.8 Schedule of Assessments

The Schedule of Assessments is presented in Table 1.

 Table 1
 Schedule of Assessments

| Period or Visit | Screenin<br>g | | | | On Tre | eatment | | | | | reatment<br>w-Up <sup>a</sup> | Premature<br>Termination | Unscheduled <sup>c</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day or Week | Day (-45)<br>to Day (-<br>1) | Day<br>1 | Wee<br>k<br>2 | Wee<br>k<br>4 | Wee<br>k<br>8 | Wee<br>k 12 | Wee<br>k 16 | Wee<br>k 20 | Wee<br>k 24 a | Week<br>28 | Week<br>36 | Varies | Varies |
| Visit Wi | ndow (days) | 0 | +/- 2 | +/- 2 | +/- 3 | +/- 3 | +/- 3 | +/- 3 | - 3 | +/- 3 | +/- 3 | N/A | N/A |
| Informed Consent(s) d | X | | | | | | | | $X^{l}$ | | | | |
| Demographic data | X | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | |
| Medication history | X | | | | | | | | | | | | |
| Liver screening e | X | | | | | | | | | | | | |
| Full physical examination | X | | | | | | | | X | | X | X | |
| 12 lead ECG | X | X | | | | X | | | X | | X | X | if indicated |
| Height and weight | X | X | | X | | | | | X | | X | | |
| Vital signs | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant medications /<br>Adverse events | | X | X | X | X | X | X | X | X | X | X | X | X |
| Confirm eligibility | | X | | | | | | | | | | | |
| Randomization (IRT) | | X | | | | | | | | | | | |
| Symptom directed physical exam | | X | X | X | X | X | X | X | | X | | | X |
| Paper diary | | X | X | X | X | X | X | X | X | | | | |
| Drug accountability | | | X | X | X | X | X | X | X | X | X j | if applicable | |
| Drug dispensation | | X | X | X | X | X | X | X | X | Х ј | | | |
| In-clinic dosing:<br>ABI-H0731/placebo | | X | X | X | X | X | X | X | X | X | | | |
| ETV dosing <sup>k</sup> | | X k | X k | X k | X | X | X | X | X | X | | | |
| Digital photography c | | | | | | | | | | | | | if indicated |
| Virology/Immunology | | | | | | | | | | | | | |
| HBV genotype | X | | | | | | | | | | | | |
| HBV viral load | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Quantitative HBsAg, quant HBeAg <sup>f</sup> | X | X | | X | X | X | X | X | X | X | X | X | X |

| HBsAb, HBeAb | X | X | | | | X | | | X | | X | X | |
|--------------|---|---|---|---|---|---|---|---|---|---|---|---|---|
| HBV RNA | X | X | X | X | X | X | X | X | X | X | X | X | X |

 Table 1
 Schedule of Assessments (continued)

| Period or Vi | it Screening | | On Treatment | | | | | | | Post-Treatment<br>Follow-Up <sup>a</sup> | | Premature<br>Termination <sup>b</sup> | Unscheduled <sup>c</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day or Wee | Day (-45)<br>to Day (-<br>1) | Day 1 | Week<br>2 | Week<br>4 | Week<br>8 | Week<br>12 | Week<br>16 | Week<br>20 | Week<br>24 a | Week<br>28 | Week<br>36 | Varies | Varies |
| HBV DNA serum resistance | | X | X | X | X | X | X | X | X | X | X | X | X |
| HIV Ab | X | | | | | | | | | | | | |
| HCV Ab; HDV Ab; HAV<br>(IgM); HEV (IgM) | X | | | | | | | | | | | | X |
| Laboratory Assessment | | | | | | | | | | | | | |
| Chemistry <sup>b</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Hematology | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Coagulation | X | X | | X | X | X | X | X | X | X | X | X | X |
| Serum AFP | X | | | | | | | | | | | | |
| FSH (females only) | X | | | | | | | | | | | | |
| Urinalysis | X | X | | X | X | X | X | X | X | X | X | X | X |
| Urine drug test | X | X | | | | | | | | | | X | X |
| Pregnancy Test g | X | X | X | X | X | X | X | X | X | X | | X | X |
| PK Sample Collection | | | | | | | | | | | | | |
| Pre-dose ABI-H0731 | | X | X | X | | X | | | X | X | | X | X |
| h ETV | | X | X | X | | X | | | X | X | | X | X |
| Optional post-dose i<br>4 (±2) hours after ABI-H0731<br>and ETV administration | | X | X | X | | | | | | | | | |
| Exploratory | | | | | | | | | | | | | |
| Optional PG sample <sup>c</sup> | | X | | | | | | | | | | | · |
| Core protein (HBCrAg) | | X | X | X | X | X | X | X | X | X | X | X | X |
| Viral nucleic acid | | X | X | X | X | X | X | X | X | X | X | X | X |

a Subjects who elect NOT to enter rollover study ABI-H0731-211 at Week 24 will discontinue ABI-H0731 and continue to take ETV during the 12-week follow-up period (inclusive of Weeks 28 and 36).

b Subjects who discontinue treatment before Week 24 should immediately undergo the assessments listed for the Premature Termination visit and then continue scheduled assessments, except that these subjects need only two further PK collections (at the Premature Termination visit and the next scheduled time point). Subjects who discontinue study assessments before completing the 12-week follow-up period should undergo the assessments listed for the Premature Termination visit.

- c Any subjects with rash or ALT flare (defined in section 4.6) should return to the clinic for an unscheduled visit as soon as possible, ideally within 3 days.
- Unscheduled visit for ALT flare: All subjects should have the laboratory findings confirmed within 3 days of receipt of the original results. All subjects should undergo a symptom directed physical examination and the following laboratory tests: ALT AST, total bilirubin, INR, and serum albumin. If the ALT flare is confirmed, perform the following tests: HBV DNA, HBV serologies (quantitative HBeAg [reflex qualitative HBeAg is negative] and HBsAg [reflex qualitative HBsAg if quantitative HBsAg is negative]), HAV IgM, HCV RNA, HDV RNA, and HEV IgM.
  - Unscheduled visit for rash: Digital photographs of the rash should be taken and blood samples should be taken (for erythrocyte sedimentation rate, complete blood count [with differential], creatinine, ALT, AST, and total bilirubin). If the rash diagnosis is uncertain, or if a rash is Grade 2, a referral to a dermatologist should be made and a biopsy should be conducted if recommended by the dermatologist. For a rash that is Grade 3 or higher, a referral to a dermatologist should be made and a biopsy should be requested of the dermatologist. All dermatologist reports and biopsy results will be included in the source and eCRF. Digital photographs of the rash should be obtained at each visit to document any change in condition. Unscheduled visits should continue until the rash has resolved or declined to Grade 1 or less for two successive visits.
- d Study specific including optional PG consent. PG sample collection requires documentation of completed PG consent.
- e Liver evaluation to be done by any protocol approved method (Biopsy, fasting FibroScan, MRI, liver ultrasound), unless a liver biopsy demonstrating lack of cirrhosis or bridging fibrosis has been conducted in the last 6 months.
- f If quantitative HBsAg or HBeAg are negative at any visit subsequent to screening, reflex to qualitative.
- A serum pregnancy test is required at screening, and on Day 1 both urine and serum should be performed (subjects may begin treatment based on urine results; any subjects negative by urine subsequently found to be positive on serum should immediately discontinue treatment and may be replaced). All post-Day 1 pregnancy tests may be conducted by urine dipstick. If positive on dipstick, please reflex to serum.
- h If the subject inadvertently administers study drug prior to collection, a PK sample should still be drawn. Refer to protocol's PK Assessments section.
- i Optional post-dose PK samples for ABI-H0731 and ETV may be collected 4 (±2) hours after in-clinic study drug + ETV administration at Day 1 and either Week 2 or Week 4. If a subject can only provide optional samples on Weeks 2 or 4, those may be collected from subjects that were not able to provide optional PK samples on Day 1.
- j Week 28 drug dispensation and Week 36 drug accountability only applies to ETV, not to ABI-H0731/placebo.
- k If subjects are not able to remain in clinic for ETV dosing, then ETV may be dosed following their clinic visit and subjects should be reminded to record the dosing time within their dosing diary.
- 1 Subjects who elect to roll over onto the open-label extension study will be required to sign a separate consent at Week 24.

Ab=antibody; AFP=alfa fetoprotein; ALT=alanine aminotransferase; AST=aspartate aminotransferase; ECG=electrocardiogram; eCRF=electronic case report form; ETV = entecavir; FSH=follicle-stimulating hormone; HAV=hepatitis A virus; HBCrAg=hepatitis B core-related antigen; HBeAb=HBeAg antibody; HBeAg=hepatitis B "e" antigen; HBsAb=HBsAg antibody; HBsAg=hepatitis B surface antigen; HBV=hepatitis B virus; HCV=hepatitis C virus; HDV=hepatitis D virus; HEV=hepatitis E virus; HIV=human immunodeficiency virus; IgM=immunoglobulin M; MRI=magnetic resonance imaging; N/A=not applicable; PG=pharmacogenomic; PK=pharmacokinetic; Quant=quantitative; ULN =upper limit of normal.

## 5 POPULATION

## 5.1 Number of Subjects

Globally, approximately 24 male or female HBeAg-positive treatment-naïve subjects with CHB, between the ages of 18 and 70, with no evidence of cirrhosis or end-stage liver disease will be randomized.

#### 5.2 Inclusion Criteria

Subjects must meet ALL of the following inclusion criteria in order to be eligible for enrollment:

- 1. Male or female between ages 18 and 70 years (inclusive)
- 2. Female subjects must agree to use dual effective birth control methods for the duration of the study and follow-up or be surgically sterile for at least 6 months or at least 2 years post-menopausal, with serum follicle-stimulating hormone (FSH) levels consistent with a post-menopausal status. Effective birth control methods include male or female condom (may not be used together due to increased risk of breakage), vasectomy, intrauterine device (IUD- including IUDs with hormonal components), diaphragm, or cervical cap. Systemic (oral/injectable) hormonal birth control are prohibited. Female subjects must have a negative serum pregnancy test at screening
- 3. All heterosexually active male subjects must agree to use dual effective birth control methods for the duration of the study and follow-up. Effective birth control methods include male or female condom (may not be used together due to increased risk of breakage), vasectomy, hormone-based contraception (only applicable to female partners of male subjects), IUD, diaphragm, or cervical cap
- 4. Body mass index (BMI) 18 to 36 kg/m<sup>2</sup> and a minimum body weight of 45 kg (inclusive)
- 5. Agreement to adhere to Lifestyle Considerations (including abstaining from alcohol abuse [defined as alcohol consumption exceeding 2 standard drinks per day on average (1 standard drink = 10 grams of alcohol)] and the use of illicit substances, herbal or other substances, or unnecessary over-the-counter medications; see Section 5.4) throughout study duration
- 6. In good general health except for chronic HBV infection (defined as HBV infection for at least 6 months documented for example by two repeated HBsAg positivity and/or history of detectable viral load documented at least two times ≥6 months apart (inclusive of screening), and serum IgM anti-HBV core-related antibody negative at screening
- 7. HBV viral load ≥2×10<sup>5</sup> IU/mL
- 8. HBeAg-positive at screening
- 9. HBsAg >1000 IU/mL at screening

# 10. Liver biopsy results of

o Metavir F0-F2 (absence of bridging fibrosis or cirrhosis) within 1 year of screening

### OR

- Fasting FibroScan ≤8 kPa within 3 months of screening (including screening visit) or other Sponsor-approved hepatic imaging study (hepatic magnetic resonance imaging [MRI], or hepatic ultrasound by an ultrasongrapher with expertise in evaluation of liver fibrosis) within 6 months of screening indicating lack of cirrhosis or advanced liver disease (F0-F2 or equivalent).
  - Subjects with an ambiguous non-invasive result, eg, a fasting FibroScan >8 kPa and  $\leq$ 10 kPa are excluded unless a biopsy within the 12 months before first visit confirms the absence of bridging fibrosis and cirrhosis. Subjects with a FibroScan >10 kPa are excluded
- 11. Have the ability to take oral medication and be willing to adhere to the ABI-H0731-202 regimen in the opinion of the Investigator
- 12. Willing and able to provide informed consent

#### 5.3 Exclusion Criteria

Subjects who meet ANY of the following exclusion criteria will not be eligible for enrollment:

- 1. Co-infection with human immunodeficiency virus (HIV), HCV, HEV, or HDV
- 2. History or evidence of hepatic decompensation (including gastrointestinal bleeding or esophageal varices) at any time prior to or at time of screening
- 3. Subject is febrile (temperature >37.5°C) at screening
- 4. Clinically significant cardiac or pulmonary disease, chronic or recurrent renal or urinary tract disease, liver disease other than HBV, endocrine disorder, autoimmune disorder, diabetes mellitus requiring treatment with insulin or hypoglycemic agents, neuromuscular, musculoskeletal, or mucocutaneous conditions requiring frequent treatment, seizure disorders requiring treatment, or other medical conditions requiring frequent medical management or pharmacologic or surgical treatment that in the opinion of the Investigator or the Sponsor makes the subject unsuitable for the study
- 5. Any prior treatment with lamivudine or telbivudine, previous treatment with an investigational agent for HBV other than ABI-H0731; or any other SOC treatment for > 4 weeks
- 6. Participation in another clinical trial of a drug or device whereby the last investigational drug/device administration is within 60 days or five half-lives prior to the first study drug administration, whichever is longer
- 7. History of persistent ethanol abuse (alcohol consumption exceeding 2 standard drinks per day on average [1 standard drink = 10 grams of alcohol]) or illicit drug abuse within 3 years before screening

- 8. Females who are lactating or pregnant or wish to become pregnant
- 9. History of HCC
- 10. A history of malignancy other than HCC unless the subject's malignancy has been in complete remission off chemotherapy and without additional medical or surgical interventions during the 3 years before screening
- 11. Previous treatment with or contraindication to use of ETV per local prescribing information
- 12. Exclusionary laboratory results
  - a. Platelet count <100,000/mm<sup>3</sup>
  - b. Albumin < LLN
  - c. Total bilirubin >1.2×ULN unless known Gilbert syndrome; subjects with Gilbert syndrome are eligible if direct bilirubin is within normal limits
  - d. Direct bilirubin >1.2×ULN
  - e. ALT >10×ULN at screening
  - f. Serum alpha fetoprotein (AFP) ≥100 ng/mL. If AFP at screening is >ULN but <100 ng/mL, subject is eligible if a hepatic imaging study prior to initiation of study drug reveals no lesions suspicious of possible HCC
  - g. Prothrombin time: INR >1.5×ULN
  - h. Glomerular filtration rate (GFR) <60 mL/min/1.73 m² by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation [Levey 2009]
  - i. Serum hemoglobin A1c (HbA1c) >8%
  - j. Any other laboratory abnormality deemed clinically significant by the Sponsor or the Investigator

### 5.4 Lifestyle Considerations

During this study, subjects are asked to:

- Abstain from abuse of alcohol (in the opinion of the Investigator; abuse is considered alcohol consumption exceeding 2 standard drinks per day on average [1 standard drink = 10 grams of alcohol]) and from any use of illicit substances for the duration of the study
- Abstain from the use of herbal or other supplements

• Abstain from use of over-the-counter concomitant medications unless they are medically indicated for the health and well-being of the subject in the opinion of the Principal Investigator

#### 5.5 Screen Failures

Screen failures are defined as subjects who consent to participate in the clinical trial but are not subsequently randomly assigned to the study intervention or entered in the study. Individuals who do not meet the criteria for participation in this trial (screen failure) because of an abnormal screening laboratory value may be rescreened one time. Rescreened subjects should be assigned the same subject number as for the initial screening.

# 5.6 Strategies for Recruitment and Retention

Approximately 24 subjects will be enrolled globally.

Subject recruitment will be performed by the study sites in accordance with local standards and regulations and be detailed in a separate plan.

Subjects who complete the treatment phase of this study will be eligible to receive open-label ABI-H0731 and ETV in an extension study.

### 6 STUDY DRUG

# 6.1 Description

ABI-H0731 active pharmaceutical ingredient (API) is manufactured under current Good Manufacturing Practices (GMP) via standard synthetic chemistry methods.

**Drug Substance** 

| Code name | ABI-H0731 |
|------------------------------|------------------|
| US Adopted Name | Not yet assigned |
| International Nonproprietary | |
| Name | Not yet assigned |
| Relative molecular mass | 467.44 amu |

**Physicochemical Properties** 

| Appearance | White to off-white powder |
|---------------|---------------------------|
| Physical form | Crystalline |
| Melting point | 301°C |

## **Solubility**

| 0.1 N HCl (pH 1.1) | 4 μg/mL |
|--------------------|------------|
| FaSSIF (pH 6.5) | 35 μg/mL |
| Acetone | 17 mg/mL |
| Dimethyl acetamide | >625 mg/mL |
| Ethanol | Insoluble |

FaSSIF=fasted state simulated intestinal fluid; HCl = hydrochloride

#### 6.1.1 Formulation

The drug product is a tablet containing ABI-H0731 in a solid dispersion produced by spray drying a solution of ABI-H0731 with an inert polymer. This spray-dried dispersion has been mixed with standard pharmaceutical excipients, such as microcrystalline cellulose, mannitol, croscarmellose sodium, and magnesium stearate, and compressed into a tablet containing approximately 100 mg ABI-H0731, manufactured according to GMP. Matching placebo tablets contain the same excipients and are also manufactured according to GMP.

#### **6.1.2 Storage**

Bottled drug product at the study site should be stored at controlled room temperature (15°C to 30°C [59°F to 89°F]) in a secure, locked location at the sites, accessible only to study personnel.

## 6.2 Packaging and Shipment

ABI-H0731 tablets and matching placebo tablets are packaged in high density polyethylene bottles fitted with child-resistant screw caps containing a desiccant (silica gel) and shipped to sites under at ambient conditions (15°C to 30°C [59°F to 89°F]).

#### 6.3 Dose and Administration

# 6.3.1 Dosing in the Study

All subjects will take ABI-H0731 or matching placebo as three 100-mg tablets once daily. Dosing should be after a meal, and at approximately the same time each day. ETV should be taken as recommended per package insert.

On study treatment visit days, ABI-H0731/placebo will be administered in the clinic; subjects will self-administer on all other treatment days. On study treatment visit days which include PK collection, subjects will administer ABI-H0731/placebo in clinic, and if possible, also the ETV in the clinic. Study personnel will document time of study drug administration in subject's medical record. Subjects will be required to record the dates and times of each dose they self-administer in a diary.

Refer to the Site Operations Manual for detailed instructions on managing missed or incorrect doses.

#### 6.3.2 Preparation

Not applicable.

### 6.3.3 Blinding

Study subjects and site personnel administering the study drug and performing the clinical assessments on the subjects, will be blinded to individual subjects' treatments assignments (ABI-H0731 + ETV therapy or placebo + ETV therapy). The DMC, as well as select individuals at the Sponsor and the CRO will not be blinded to subjects' treatment assignments to facilitate randomization, prompt analysis of any arising safety/tolerance issues, and the Week 12 safety data review. As this is an exploratory Phase 2a study, certain individuals may also be unblinded to the efficacy results before the final analysis.

### 6.4 Accountability

Regulatory requirements stipulate accounting of all investigational drug received by the study site. Records of drug disposition must include the date received by the site, date administered, quantity administered, and the subject to whom study drug was administered. The Investigator is responsible for the accountability of all used and unused study drug containers and unused study drug.

The study site is to use a study drug accountability record to document study drug disposition. All items on this form are to be fully completed. The Sponsor or the CRO will confirm if the method of recording study drug accountability by the clinical site and the location of study drug records at the site is appropriate.

Each time study personnel dispense study drug for a subject, he or she is to record the date dispensed, the number of tablets or vials of study drug dispensed, and his or her initials. Study site personnel are to monitor the inventory of clinical supplies and maintain a count of all used and unused containers. The clinical monitor will review study drug and ETV accountability records during monitoring visits. The site pharmacist or designated staff member will keep accurate records of drug dispensation routinely during the study. Study drug and ETV dispensation is planned for Day 1 and each scheduled visit thereafter during the dosing period.

## 6.5 Compliance

To monitor compliance and to facilitate drug accountability at the study site, subjects will be required to record each dose they take in a diary. Subjects will also be asked to return used bottles and any unused study drug at study visits. Subjects who forget to return bottles will be asked to return them at the next study visit.

# 6.6 Concomitant Therapy

A concomitant medication is defined as any prescription or over-the-counter preparation, including vitamins, over-the-counter medications, and supplements. For all randomized subjects, all concomitant medications are discouraged, and any concomitant medications must be recorded in the designated eCRF from the date informed consent is obtained to 30 days following the last dose of all study drug(s).

All subjects on this study will initiate and continue ETV for the duration of the study. Subjects will provide a log of their ETV therapy together with that of ABI-H0731/placebo at each clinic visit.

### 6.6.1 Prohibited Concomitant Therapy

As the potential for drug-drug interactions between ABI-H0731 and other compounds has not yet been fully evaluated, consumption of grapefruit/grapefruit juice is forbidden. Systemic (oral, injectable or implanted) hormonal birth control is not permitted as an acceptable means of birth control for female subjects of child bearing potential. Additional prescription medication use is discouraged, unless required for an emergent medical need occurring during the course of the study. To the extent possible, medications with narrow therapeutic indices should be avoided. In particular, medications metabolized by cytochrome P450 (CYP) isoenzymes 2B6, 2C8, 2C9, or 2D6 should be avoided (see APPENDIX III). Concomitant prescription medications, over-the-counter medications, and supplements will be reported in the eCRF.

#### 6.6.2 Other Medications and Treatments

Within the suggested guidelines above, subjects may receive any other medication or treatment that is deemed medically necessary by the Study Investigator. All medication and treatments should be recorded in the eCRF, including name of the medication or treatment, the start and stop dates, and the indication.

# 7 STUDY CONDUCT

# 7.1 Study Procedures by Time Point

Refer to the Schedule of Assessments (Table 1).

#### 7.2 Discontinuation

### 7.2.1 Discontinuation from Treatment

If an individual study participant is not satisfactorily tolerating study drug treatment in the judgment of the clinical investigator, then – in consultation with the Sponsor - that participant may be discontinued from treatment. Discontinuation from treatment does not mean discontinuation from the study. Subjects who discontinue treatment before Week 24 should immediately undergo the assessments listed for the Premature Termination visit (Table 1) and then continue scheduled assessments, except that these subjects need only two further PK collections (at the Premature Termination and the next scheduled time point). If a clinically significant finding is identified (including, but not limited to changes from Baseline) after enrollment, the Investigator or qualified designee will determine if any change in subject management is needed. Any new clinically relevant finding will be reported as an adverse event.

In this study, subjects will be closely monitored for any evidence of worsening hepatic function or evidence of dermatologic adverse events. Subjects with post-Baseline ALT elevations of 2-fold or higher will be closely monitored. Study treatment will be discontinued in subjects with confirmed evidence of declining hepatic function during treatment (Section 4.6.1).

Specific guidance on management and the data to be collected at the time of study intervention discontinuation are described below.

Any subjects negative by urine pregnancy test on Day 1 who are subsequently found to be positive on serum pregnancy test should immediately discontinue treatment and may be replaced.

## 7.2.2 Discontinuation from Study

Discontinuation from study (withdrawal of consent) means that the subject does not wish to receive further protocol-required therapies or undergo protocol-required procedures, and the subject does not wish to or is unable to continue further study participation. Subjects who discontinue during follow-up should undergo the assessments listed for the Premature Termination visit unless they withdraw consent to do so. Subject data up to withdrawal of consent will be included in the analysis of the study, and where permitted, publicly available data can be included after withdrawal of consent. The Investigator is to discuss with the subject appropriate procedures for withdrawal from the study.

# 8 DESCRIPTION OF STUDY PROCEDURES

# 8.1 Efficacy Assessments

To provide an assessment of the antiviral efficacy of ABI-H0731 in treatment-naïve HBV subjects, this study will evaluate treatment-related changes in serum viral DNA, serum HBsAg, serum HBeAg, HBCrAg, and serum HBV RNA levels. Additionally, in CHB subjects where HBV DNA is detectable is serum, an evaluation will be made to determine if HBV has become undetectable.

To assure standardization of the virologic methods in this study, HBV DNA-related and HBV antigenrelated virologic assessments will be conducted at a central reference laboratory. Subject serum samples for resistance-related sequencing and HBV RNA testing will be shipped frozen to the Sponsor or a designated third-party laboratory for testing.

# 8.1.1 Primary Efficacy Assessment

The primary endpoint is change in mean  $\log_{10}$  HBV DNA from Baseline (Day 1) to Week 12 or Week 24 on ABI-H0731 + ETV as compared to placebo + ETV. Samples for quantitative HBV DNA levels will be collected at screening, Day 1, and Weeks 2, 4, 8, 12, 16, 20, and 24 (or at the time of discontinuation). Follow-up samples will be collected Weeks 28 and 36 for subjects who do not continue treatment in the extension protocol. Subjects who enter the continuation protocol will have samples collected according to the extension protocol.

# 8.1.2 Secondary and Exploratory Efficacy Assessments

Blood samples for the assessment of secondary and exploratory efficacy endpoints will be collected as described below. For all analytes, the follow-up samples will only be collected for subjects who do not continue treatment in the extension protocol. Subjects will have the following samples collected according to the Schedule of Assessments (Table 1).

- Quantitative/qualitative HBsAg and HBeAg levels
- HBsAb and HBeAb
- HBV RNA
- HBCrAg (HBV Core related Antigen)
- HBV resistance samples
- Samples for exploratory viral research

### 8.2 Safety Assessments

For adverse events, see Section 9.

For serious adverse events, see Section 10.

# 8.2.1 Clinical Laboratory Tests

Clinical laboratory tests will be performed at the timepoints indicated in the Schedule of Assessments (Table 1). The clinical laboratory assessments are listed in Table 2.

**Table 2** Clinical Laboratory Tests

| Panel | Tests |
|---|---|
| Clinical chemistries | Blood glucose levels, serum or plasma electrolytes (sodium, potassium, chloride, bicarbonate), calcium, blood urea nitrogen, creatinine, uric acid, total and direct bilirubin a, ALT, AST, GGT, alkaline phosphatase, LDH, amylase, triglycerides, total cholesterol, inorganic phosphate or total phosphate, total protein, albumin, lipase, and total serum or plasma globulins |
| In case of ALT flares | ALT, AST, total bilirubin, serum albumin, and INR |
| Hematology | Complete blood counts: hemoglobin, hematocrit, RBC indices (MCV, MCHC), reticulocyte counts, leukocyte counts (total and differential), and platelet counts |
| Coagulation | Prothrombin time/INR and aPTT |
| Urinalysis | pH, specific gravity, protein, glucose, ketones, and occult blood |
| Other | AFP, HbA1c, and FSH |
| Pregnancy tests | For females only; a serum or plasma pregnancy test must be performed at screening, and both serum/plasma and urine are required Day 1; a serum, plasma, or urine pregnancy test must be performed at all subsequent visits. A positive result disqualifies the subject for study treatment |
| Urine drug screening | Amphetamine/methamphetamine, barbiturates, benzodiazepines, cannabinoids, cocaine metabolite, ecstasy, ethanol, opiates, phencyclidine, and propoxyphene. Note: If cannabinoids are not illegal in the subject's local, cannabinoids are not exclusionary |
| Antibodies | HCV, HDV, HAV IgM, HEV IgM, and HIV |

AFP=alpha fetoprotein; ALT=alanine aminotransferase; aPTT=activated partial thromboplastin time; AST=aspartate aminotransferase; FSH=follicle-stimulating hormone; GGT=gamma-glutamyl transpeptidase; HAV=hepatitis A virus; HbA1c=hemoglobin A1c; HCV=hepatitis C virus; HDV=hepatitis D virus; HEV=hepatitis E virus; HIV=human immunodeficiency virus; IgM=immunoglobulin M; INR=International Normalized Ratio; LDH=lactate dehydrogenase; MCHC=mean corpuscular hemoglobin concentration; MCV=mean corpuscular volume; RBC=red blood cell; ULN=upper limit of normal

a Perform fractionated bilirubin, if total bilirubin >ULN.

During the study, any clinically significant laboratory abnormality or clinically significant change from Baseline should be recorded as an adverse event (Section 9).

# 8.2.2 Other Safety Assessments

Other safety assessments include the following:

Vital signs.

- Twelve-lead ECG. During the study, any clinically significant ECG result or change from Baseline should be confirmed, and if confirmed, should be recorded as an adverse event (Section 9).
- Concomitant medications, including supplements and over-the-counter medications, will be recorded.

#### **8.3** Pharmacokinetic Assessments

Pre-dose samples will be collected to determine trough concentrations of ABI-H0731 and ETV. Post-dose samples for both ABI-H0731 and ETV will be collected from subjects willing and able to provide the optional sample  $4 \pm 2$  hours after dosing. Sample timing is outlined in Table 3.

**Table 3** Pharmacokinetic Sample Collection

| Time Period | Timepoint <sup>a</sup> | Time Relative to Study Drug<br>Administration <sup>b</sup> |
|---|---|---|
| | Study Day 1 pre-dose | Before |
| Double-blind | Study Weeks 2, 4, 12, 24 predose | Before |
| Treatment | OPTIONAL <sup>c</sup> Day 1, Week 2, and/or Week 4, post-dose (see laboratory manual) | 4 (±2) hours post-dose |
| Follow-up | Study Week 28 pre-dose | Collect at same time with other central labs |

- a A pharmacokinetic sample should be collected if an unscheduled or early termination visit is performed.
- b Sample collection times are targeted times. Samples collected outside of these targeted times will not be considered protocol deviations as long as the actual time the sample is collected is accurately recorded on source documentation and the case report form.
- c If a subject can only provide optional samples on Weeks 2 or 4, those may be collected from subjects that were not able to provide optional pharmacokinetic samples on Day 1.

### 8.4 Other Assessments

Other assessments include the following:

Liver assessment at screening: To be eligible, subjects must have liver biopsy results of

Metavir F0-F2 (absence of bridging fibrosis or cirrhosis) within 1 year of screening

#### **OR**

○ Fasting FibroScan ≤8 kPa within 3 months of screening (including screening visit) or other Sponsor-approved hepatic imaging study (hepatic MRI, or hepatic ultrasound by a ultrasongrapher with expertise in evaluation of liver fibrosis) within 6 months of screening indicating lack of cirrhosis or advanced liver disease (F0-F2 or equivalent). FibroScan should be conducted after an overnight fast.

Subjects with an ambiguous non-invasive result, eg, a fasting FibroScan >8 kPa and  $\leq$ 10 kPa are excluded unless a biopsy within the 12 months before first visit confirms the absence of bridging fibrosis and cirrhosis. Subjects with a FibroScan >10 kPa are excluded.

Demography, medical history, and full physical examination will be performed at screening.

Pharmacogenomic samples will be collected at Day 1 for subjects who consent to this procedure. These samples may be saved for future research.

### **8.5** Protocol Deviations

Any deviations from the protocol will be identified by the site monitor, medical monitor, site staff, or statistician, based on the protocol and criteria defined in the Medical Monitoring Plan. Identified deviations will be confirmed and documented by the site monitor. Prior to database lock, protocol deviations will be reviewed and a list of important protocol deviations, and subjects who will be excluded from the per-protocol (PP) dataset will be determined based on blinded review of data.

# 9 ADVERSE EVENTS

An adverse event is any untoward medical occurrence in a study subject administered an investigational product(s) regardless of the causal relationship with treatment.

An adverse event, therefore, can be any unfavorable and unintended sign (including laboratory finding), symptom, or disease temporally associated with participation in an investigational study, whether or not considered drug related. In addition to new events, any increase in the severity or frequency of a pre-existing condition that occurs after the subject signs the Informed Consent Form (ICF) for participation is considered an adverse event. This includes any side effect, injury, toxicity, or sensitivity reaction.

# 9.1 Documenting Adverse Events

Adverse events will be monitored throughout the entire study. Investigators will ask the subject at each visit if they have experienced any untoward effects since the last study visit. All adverse events will be recorded on the eCRFs provided: a description of the event, severity, time of occurrence, duration, any action (eg, treatment and follow-up tests), and the outcome should be provided along with the Investigator's assessment of the relationship to the study treatment.

Adverse events will be recorded from the time written informed consent is signed until completion of the Week 36 follow-up visit or until 30 days following cessation of the last dose of treatment with the study drug for subjects who discontinue from follow-up.

# 9.2 Assessment of Intensity

The severity of each adverse event and laboratory abnormality is to be assessed by the Investigator according to the modified Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events (APPENDIX II), which grades the severity of clinical adverse events and laboratory abnormalities in a four-category system.

For adverse events not included in APPENDIX II, the following guidelines will be used to describe severity:

- Mild (Grade 1): Mild symptoms causing no or minimal interference with usual social & functional activities with intervention not indicated
- Moderate (Grade 2): Moderate symptoms causing greater than minimal interference with usual social & functional activities with intervention indicated
- Severe (Grade 3): Severe symptoms causing inability to perform usual social & functional activities with intervention or hospitalization indicated (Of note, the term "severe" does not necessarily equate to "serious")
- Life-Threatening (Grade 4): Potentially life-threatening symptoms causing inability to perform basic self-care functions with intervention indicated to prevent permanent impairment, persistent disability, or death

Note that an adverse event or laboratory abnormality that is life-threatening as it exists constitutes a serious adverse event.

# 9.3 Assessment of Causality

All adverse events must have their relationship to study intervention assessed by the clinician who examines and evaluates the subject based on temporal relationship and his/her clinical judgment. Each adverse event must be recorded in the source and eCRF, whether serious or not serious. For the purposes of this study each event is to be assessed with regard to the following causality categorizations, in the Investigator's considered judgment:

- **Not related**: An adverse event with sufficient evidence to accept that there was no causal relationship to administration of study medication (eg, no temporal relationship because the study medication was administered after the onset of the event, an investigation showed that study medication was not administered, another cause was proven).
- Unlikely related: An adverse event, including a clinical laboratory test abnormality, with a temporal relationship to administration of study medication that made a causal relationship improbable and in which other drugs, events, or underlying disease provided plausible explanations.
- **Possibly related**: An adverse event with a reasonable time sequence to administration of study medication but that could also be explained by concurrent disease or other drugs or events. Information on drug withdrawal may have been lacking or unclear.
- **Related**: An adverse event occurred in a plausible time relationship to administration of study medication and that could not be explained by a concurrent disease or other drugs or events. The response to withdrawal of the drug (dechallenge) was clinically reasonable.

### 9.4 Expectedness

An adverse event is considered "unexpected" if it is not listed in the IB or is not listed at the specificity or severity that has been observed. The CRO and Sponsor medical monitors will be responsible for determining whether an adverse event is expected or unexpected.

### 9.5 Adverse Events of Special Interest

Adverse events of Special Interest include rash and ALT flare and should be reported using the Adverse Events form of the eCRF. There are no expedited reporting requirements for adverse events of Special Interest (other than those that meet other reporting requirements).

### 9.6 Clinical Laboratory Changes

In the event of abnormal laboratory test values, the tests should be repeated immediately. If the Investigator considers the abnormality to be clinically significant, it should be reported as an adverse event and followed up until it returns to the normal range and/or an adequate explanation of the abnormality is found.

# 9.7 Adverse Event Follow-up

After the initial adverse event or serious adverse event report, the Investigator will follow-up proactively on each subject and provide further information to the CRO on the subject's condition. During the study, all adverse events or serious adverse events should be followed up to resolution unless the event is considered by the Investigator to be unlikely to resolve due to the subject's underlying disease, or the subject is lost to follow-up.

### 9.8 Pregnancy

Pregnancy in itself is not regarded as an adverse event unless there is a suspicion that an investigational product may have interfered with the effectiveness of a contraceptive medication. However, the outcome of all pregnancies (spontaneous miscarriage, elective termination, normal birth, or congenital abnormality) must be followed up and documented even if the subject was discontinued from the study. All pregnancies must be reported using the Pregnancy Report Form within 24 hours of learning of the pregnancy following the same procedures as for reporting serious adverse events (see Section 10.2).

All reports of congenital abnormalities/birth defects are serious adverse events. Spontaneous miscarriages should also be reported and handled as serious adverse events. Elective abortions without complications should not be handled as adverse events. All outcomes of pregnancy must be reported to the CRO.

Pregnancies among female partners of male subjects will also be reported and followed for outcome.

### 10 SERIOUS ADVERSE EVENT

#### 10.1 Definition of Serious Adverse Event

A serious adverse event is any event that meets any of the following criteria:

- Death
- Life-threatening
- Inpatient hospitalization or prolongation of existing hospitalization
- Persistent or significant disability/incapacity
- Congenital anomaly/birth defect in the offspring of a subject who received ABI-H0731
- Other: Important medical events that may not result in death, be life-threatening, or require hospitalization, may be considered a serious adverse event when, based upon appropriate medical judgment, they may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such events are:
  - o Intensive treatment in an emergency room or at home for allergic bronchospasm
  - o Blood dyscrasias or convulsions that do not result in inpatient hospitalization
  - Development of drug dependency or drug abuse

#### **Definition of Terms**

Life-threatening: An adverse event is life-threatening if the subject was at immediate risk of death from the event as it occurred; ie, it does not include a reaction that if it had occurred in a more serious form might have caused death. For example, drug induced hepatitis that resolved without evidence of hepatic failure would not be considered life-threatening even though drug induced hepatitis can be fatal.

Hospitalization: adverse events requiring hospitalization should be considered serious adverse events. Hospitalization for elective surgery or routine clinical procedures that are not the result of adverse event (eg, elective surgery for a pre-existing condition that has not worsened) need not be considered adverse events or serious adverse events. If anything untoward is reported during the procedure, that occurrence must be reported as an adverse event, either "serious" or "non-serious" according to the usual criteria.

In general, hospitalization signifies that the subject has been detained (usually involving at least an overnight stay) at the hospital or emergency ward for observation and/or treatment that would not have been appropriate in the physician's office or outpatient setting. When in doubt as to whether "hospitalization" occurred or was necessary, the adverse event should be considered serious.

Disability/incapacitating: An adverse event is incapacitating or disabling if the experience results in a substantial and/or permanent disruption of the subject's ability to carry out normal life functions.

### 10.2 Reporting Serious Adverse Events

All serious adverse events must be reported within 24 hours of learning about the event. This can be done by emailing or faxing a completed Safety Report Form or by direct telephone communication to the numbers below. A Safety Report Form must follow all telephone reports within 24 hours.

## Fax, phone, or email information to the CRO:



The initial report should be promptly followed by detailed, written reports, which will include copies of relevant hospital case reports, autopsy reports, and other documents when requested and applicable. This additional information will be requested, if necessary, by the responsible monitor within 5 days of receipt of the alert report. This is to ensure that the initial reporting of serious adverse events is made to the Health Authorities within the required time period.

For a follow-up report to the authorities, the monitor may be required to collect further information for a final evaluation of the case. Reporting to the respective country Health Authorities will be the responsibility of the Sponsor and the CRO.

The CRO will be responsible for informing all central Institutional Review Boards (IRBs)/ Independent Ethics Committees (IECs) of serious adverse events as required. It will be the responsibility of the individual Investigators to inform any local IRBs/IECs of serious adverse events as required. Correspondence with the IRB(s)/IEC(s) relating to the reporting of serious adverse events will be retained in the study file.

During this trial, an SAE with onset during follow-on treatment with regulatory-approved HBV products, that is considered by the clinical investigator to be related to the use of these products, and the nature and severity of which is clearly "expected" on the basis of the regulatory-approved labels for the implicated product, will not be reported to regulatory authorities in an expedited manner, but will be included in the periodic safety reviews by the Sponsor and DMC for this study. Such SAEs will also be included in all data summaries submitted to national regulatory bodies and ECs/IRBs, and will be included in the eventual clinical study report.

### 10.3 Overdose

An overdose is defined as the accidental or intentional administration of any dose of a product that is considered both excessive and medically important. An overdose is not in and of itself considered to be an adverse event unless it results in untoward medical effects. Any adverse event associated with an overdose or incorrect administration of study drug should be recorded on the Adverse Event eCRF. If the associated adverse event fulfills the criteria of a serious adverse event, then the event should be reported to the Sponsor or CRO within 24 hours after the site learns of the event.

### 11 STATISTICS

# 11.1 Statistical Hypotheses

As a proof-of-concept trial, there are no statistical hypotheses, per se, regarding treatment effects in this study. Rather, displays and comparisons of study results, regarding dose-related safety, efficacy, and PK profiles among the treatment groups, will primarily utilize descriptive statistics, as noted below.

### 11.2 Sample Size

The primary objective of the study will be measured by changes from Baseline to Week 12 or Week 24 in mean  $log_{10}$  HBV DNA. As the results for this study will be used to collect information for future studies, both timepoints will be reviewed independently, with no control of the alpha level.

With a sample size of 24 subjects, randomized in a 1:1 ratio (12 active:12 placebo), a 2-sample t-test test for mean difference with a 2-sided 0.05 significance level has 87.7% power to detect a difference of at least 0.4 log<sub>10</sub> (IU/mL) in the change from Baseline in serum HBV DNA level at Week 12 or Week 24 between the placebo + ETV and ABI-H0731 + ETV groups, where an equal standard deviation of 0.3 is assumed for both groups (Table 4).

Table 4 Power Calculations under Various Mean Differences in the Change from Baseline in HBV DNA levels at Week 12 or 24 between Treatment Groups

| | Power for N=24 subjects<br>(12 ABI-H0731 + ETV: 12 Placebo + ETV) | | | |
|---|---|---|---|---|
| Estimated mean difference at Week 12<br>or Week 24 between placebo + ETV<br>and ABI-H0731 + ETV groups change<br>from Baseline HBV DNA levels | SD = 0.25 | SD = 0.30 | SD = 0.50 | SD = 0.60 |
| 0.25 log <sub>10</sub> IU/mL | 0.649 | 0.497 | 0.216 | 0.164 |
| 0.30 log <sub>10</sub> IU/mL | 0.802 | 0.649 | 0.290 | 0.216 |
| 0.40 log <sub>10</sub> IU/mL | 0.963 | 0.877 | 0.466 | 0.346 |
| 0.50 log <sub>10</sub> IU/mL | 0.997 | 0.974 | 0.649 | 0.497 |
| 0.60 log <sub>10</sub> IU/mL | >0.999 | 0.997 | 0.802 | 0.649 |

Calculated using SAS, based on a two-sided, two-sample t-test for mean differences, assuming equal weight of treatment groups, and alpha=0.05.

ETV=entecavir; HBV=hepatitis B virus; SD=standard deviation

#### 11.3 Analysis Populations

The following populations for analysis will be used in this study:

Intent-to-treat (ITT) Population: The ITT population will be defined as all randomized subjects. Subjects in this population will be analyzed according to their randomized treatment assignment, regardless of the actual treatment received.

Per-Protocol (PP) Population: The PP population will include subjects who are at least 80% compliant with scheduled study drug dosing in the 24-week treatment period, and who have no major protocol violations.

Safety Population: The safety population will include all randomized subjects who received at least one dose of study drug. Subjects in this population will be analyzed according to the actual treatment received.

Pharmacokinetic (PK1) Population 1: The PK1 population will include all subjects in the safety population who have ABI-H0731 PK data assessments available.

Pharmacokinetic (PK2) Population 2: The PK2 population will include all subjects in the safety population who have ETV PK data assessments available.

Additional populations may be defined in the statistical analysis plan (SAP).

#### 11.4 Statistical Methods

#### 11.4.1 General Considerations

Information regarding the safety, PK, and efficacy analyses is given below. An SAP containing the detailed planned statistical methods will be finalized prior to locking of the study database for the analyses, and it will form the basis for the programming of the displays and analyses of the final study data. The plan will define populations to be used for each analysis endpoint, outline all data handling conventions including missing data methods, and specify statistical methodology to be used for analysis of safety and efficacy.

Subgroup analyses will be conducted to assess virologic efficacy endpoints in subjects infected with different HBV genotypes and for subject subgroups with different baseline characteristics which could potentially influence the efficacy, safety, or PK observations in this study, eg, pre-treatment ALT level, HBsAg level, HBeAg level, ethnicity, gender, etc. These and other subgroup analyses will be further defined in the SAP.

#### 11.4.2 Primary Endpoint(s)

The primary endpoint is change in mean  $log_{10}$  HBV DNA from Baseline (Day 1) to Week 12 or Week 24 on ABI-H0731 + ETV as compared to placebo + ETV. The primary comparison will be made using a two-sided, two-sample t-test for mean differences with alpha=0.05.

### 11.4.3 Secondary and Exploratory Endpoint(s)

Secondary and exploratory endpoints will be analyzed descriptively. All secondary and exploratory efficacy endpoints will be summarized (Section 3.2.2 and Section 3.2.3).

For continuous variables, such as observed and change from Baseline HBV DNA values at each timepoint, descriptive statistics will be used, and will include the number, mean, standard deviation, median, minimum, maximum, and interquartile range and, where appropriate, a 95% CI. Missing data

methods and imputation rules will be defined in the SAP. Additional sensitivity analysis may also be performed and will be described in the study SAP.

For categorical variables, such as subjects with a 1 log<sub>10</sub> drop in serum HBsAg or HBeAg titers from Baseline and subjects with HBeAg (and HBsAg) loss and seroconversion, descriptive statistics will include number and percent who meet the endpoint criteria.

Kaplan-Meier methods will be used to evaluate time to event variables (eg, time to HBsAg loss), and the treatment groups will be compared using log-rank tests.

Cox proportional hazards regression models will be used to identify baseline factors associated with HBsAg loss rates, as defined in the SAP.

Descriptive p-values may be defined in the SAP.

## 11.4.4 Pharmacokinetic Endpoints and Analyses

The following will be analyzed descriptively:

- Trough levels and (for subjects who provide optional post-dose samples) trough to peak ratios of ABI-H0731 on ABI-H0731 + ETV therapy
- Trough levels and (for subjects who provide optional post-dose samples) trough to peak ratios of ETV on ABI-H0731 + ETV therapy as compared with placebo + ETV therapy

After all subjects have completed Week 4 (or discontinued before completing Week 4), PK data will be reviewed by an unblinded pharmacology reviewer to ensure ETV steady-state PK levels are not being affected by combination treatment with ABI-H0731. All PK time points will be included in the final analysis.

## 11.4.5 Analysis of Safety

The safety parameters to be assessed are described in Section 8.2, Section 9, and Section 10. Displays for safety results will utilize descriptive statistics. No formal hypothesis testing of safety data is planned; however, exploratory p-values to assess any potential treatment-related differences in the incidence of clinical adverse events, laboratory abnormalities, and treatment-emergent abnormal ECGs may be defined in the SAP.

Adverse events summaries will be tabulated by Medical Dictionary for Regulatory Activities (MedDRA) body system and preferred term, for each treatment group. Summaries will include all adverse events, adverse events considered possibly or probably related to treatment, Grade ≥3 (or severe) adverse events, and serious adverse events. All adverse events will be listed by subject. Any adverse events leading to premature discontinuation from the study intervention and serious treatment-emergent adverse events will be presented as a separate table or a listing.

Clinical laboratory results will be summarized descriptively by treatment group including values, changes from Baseline, and incidence of laboratory abnormalities. Laboratory results will be listed for each subject.

Exposure to treatment will be summarized descriptively, and compliance on treatments for both active and placebo (matching ABI-H0731 100-mg tablets) will be evaluated.

Vital sign data reported at each visit will be displayed by treatment, using descriptive statistics for observed and change from Baseline values.

Any post-screening changes in physical examination findings will be summarized in tabular form, by treatment group.

# 11.4.6 Demographic and Baseline Characteristics

Other variables, including subject disposition and demographic and baseline characteristics will be summarized descriptively by treatment group. The demographics and baseline characteristics include age (in years, at time of signing informed consent), race, ethnicity, height, weight, BMI, HBV genotype, and pre-treatment ALT levels.

### 11.5 Interim Analysis

No formal interim analyses are planned. See Section 12.2 for the Week 12 safety analysis and Section 8.3 for the Week 4 PK analysis.

#### 11.6 Exploratory Analyses

Multiple exploratory endpoints may be assessed in this study. NUCs of the HBV Pol/RT inhibit HBV DNA synthesis from encapsidated pre-genomic HBV RNA, resulting in reductions in serum HBV DNA levels. In NUC-treated subjects, while circulating HBV DNA declines due to inhibition of HBV Pol/RT activity, encapsidated HBV RNA remains detectable in circulating virus particles. This is not seen with CpAMs such as ABI-H0731 because the mechanisms of action by which viral load is reduced with ABI-H0731 differs from that of NUCs. As an HBV CpAM, ABI-H0731 specifically induces accelerated misassembly of HBV core protein into oligomers, with reduced incorporation of pre-genomic HBV RNA into functional nucleocapsids. In contrast to HBV NUC therapies, ABI-H0731 treatment may reduce circulating levels of HBV RNA [Wang 2016]. By altering the encapsidation and tertiary structure of HBV capsid, ABI-H0731 may potentially reduce circulating HBCrAg. When ETV is used in conjunction with a CpAM, inhibition of multiple aspects of the viral life cycle may also lead to accelerated loss of viral cccDNA.

Analysis of changes in serum HBV DNA, HBV antigen kinetics, viral RNA and HBCrAg levels in this study may thus provide additional assessments of antiviral efficacy and unique mechanisms of ABI-H0731 in HBV subjects.

Data collected for this study will be analyzed and stored by the CRO. After the study is completed, the de-identified, archived data will be stored by the Sponsor or their designee.

With the participant's approval and as approved by local IRBs/IECs, de-identified biological samples will be stored by the Sponsor or their designee. These samples could be used to research CHB, its complications and other conditions for which individuals with CHB are at increased risk, and to improve treatment. The Sponsor will also have a code-link that will allow linking the biological specimens with the phenotypic data from each participant, maintaining the blinding of the identity of the participant.

### 12 ETHICS AND RESPONSIBILITIES

#### 12.1 Good Clinical Practice

This study will be conducted in compliance with IRB/IEC and International Council for Harmonisation (ICH) Good Clinical Practice (GCP) Guidelines; Title 21 Part 56 of the US Code of Federal Regulations (CFR) relating to IRBs/IECs and GCP as described in the US FDA CFR (21 CFR § 50, 56, 312; applicable ICH guidelines regarding clinical safety data management (E2A, E2B(R3)); European Community directives 2001/20, 2001/83, 2003/94 and 2005/28 as enacted into local law, and with ICH guidelines regarding scientific integrity (E4, E8, E9, and E10). In addition, this study will adhere to all local regulatory requirements, and requirements for data protection.

## 12.2 Data Monitoring Committee

A DMC external to the Sponsor and the CRO will be formed with members consisting of individuals chosen for their expertise in treatment of HBV. Members of the DMC will include, at a minimum, physicians external to the Sponsor and the CRO and appropriate statistical representation. The primary role of this independent DMC will be to monitor safety data.

The DMC will review unblinded safety data at specified intervals, including the Week 12 safety data (Section 11.5), as outlined in the DMC charter.

In addition, the DMC will communicate major safety concerns and recommendations regarding study modification or termination to the Sponsor senior management at any time during the conduct of the study.

Records of all DMC decisions will be archived by the CRO. Selected Sponsor or their designees may serve as liaisons with the external DMC, but will not be voting members, and will not be unblinded to the results. Details regarding the DMC will be provided in the DMC charter.

### 12.3 Institutional Review Board/Independent Ethics Committee

Before initiating a trial/study, the Investigator/institution must have written and dated approval/favorable opinion from the IRB/IEC for the study protocol/amendment(s), written ICF, any consent form updates, subject recruitment procedures (eg, advertisements), and any written information to be provided to subjects and a statement from the IRB/IEC that they comply with GCP requirements. The IRB/IEC approval must identify the protocol version as well as the documents reviewed.

#### 12.4 Informed Consent

The Investigator will explain the benefits and risks of participation in the study to each subject or the subject's legally acceptable representative and obtain written informed consent. Written informed consent must be obtained prior to the subject entering the study and before initiation of any study-related procedure (including administration of investigational product).

The Sponsor or its designee will provide a sample ICF. The final, version dated, ICF must be agreed to by the Sponsor and the IRB/IEC and will contain all elements in the sample form, in language readily understood by the subject. Each subject's original consent form must be personally signed and dated by the subject or by the subject's legally acceptable representative, and by the person who conducted the informed consent discussion. The original, signed ICF will be retained by the Investigator. The Investigator will supply all enrolled subjects with a copy of their signed ICF.

The ICF may need to be revised during the study should important new information become available that may be relevant to the safety of the subject. In this instance approval should always be given by the IRB/IEC and existing subjects informed of the changes and reconsented. This is documented in the same way as previously described.

The Investigator should encourage subjects to inform their primary physician about their participation in the clinical study.

# 12.5 Records Management

#### 12.5.1 Source Documentation

Source documents contain the results of original observations and activities of a clinical investigation. Source documents include, but are not limited to, medical records (progress notes), computer printouts, screening logs, and recorded data from automated instruments.

All source documents from this study will be maintained by the Investigator and made available for inspection by authorized persons. The original signed informed consent for each subject shall be filed with records kept by the Investigator and a copy shall be given to the subject.

### 12.5.2 Study Files and Record Retention

Records must be retained in accordance with the current ICH guidelines on GCP. All essential study documents including records of subjects, source documents, eCRFs, and investigational product inventory must be kept on file.

Essential documents should be retained until at least 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region, or until at least 2 years have elapsed since the formal discontinuation of clinical development of the investigational products. However, essential documents may be retained for a longer period if required by the applicable regulatory requirements or by agreement with the Sponsor. The Sponsor is responsible for informing the Investigator when these documents need no longer be retained.

The Investigator will not dispose of any records relevant to this study without written permission from the Sponsor and will give the Sponsor the opportunity to collect such records. The Investigator shall take responsibility for maintaining adequate and accurate hard copy source documents of all observations and data generated during this study. Such documentation is subject to inspection by the Sponsor, its representatives, and regulatory authorities.

If an Investigator moves, withdraws from an investigation, or retires, responsibility for maintaining the records may be transferred to another person who will accept responsibility. Notice of transfer must be made to and agreed by the Sponsor.

### 12.6 Conflicts of Interest

Any conflict of interest of persons who have a role in the design, conduct, analysis, publication, or any aspect of this trial will be disclosed and managed. Furthermore, persons who have a perceived conflict of interest will be required to have such conflicts managed in a way that is appropriate to their participation in the design and conduct of this trial.

# 13 DATA MANAGEMENT, AUDITING, AND MONITORING

# 13.1 Data Management

An eCRF will be used for the current study, and a data management plan will be prepared by the CRO. The data will be collected via electronic data capture (EDC) using the eCRFs. The site will be responsible for data entry into the EDC system. In the event of discrepant data, the CRO will request data clarification from the sites, which the sites will resolve electronically in the EDC system. The CRO will be responsible for the data management of this trial, including quality checking of the data.

The data management methodology will be consistent with the CRO's standard operating procedures and applicable regulatory guidelines. The data management plan will specify methods to ensure the accuracy and quality of the study data.

Previous and concomitant medications will be coded using the latest available WHO Drug Reference Dictionary. Coexistent diseases and adverse events will be coded using MedDRA.

When the database has been declared to be complete and accurate, the database will be locked. Any changes to the database after that time can only be made by written agreement between the Sponsor (or designee) and the CRO project team.

## 13.2 Auditing

The Sponsor or their designed, the CRO, may conduct audits at the investigative sites including, but not limited to, drug supply, presence of required documents, the informed consent process, and comparison of eCRFs with source documents. All medical records (progress notes) must be available for audit. The Investigator agrees to participate with audits conducted at a convenient time in a reasonable manner.

Government regulatory authorities may also inspect the site during or after the study. The Investigator or designee should contact the Sponsor or the CRO, immediately if this occurs. The site must cooperate fully with regulatory authorities or other audits conducted at a convenient time in a reasonable manner.

The purpose of an audit is to assess whether ethical, regulatory, and quality requirements are fulfilled.

## 13.3 Monitoring

The Sponsor or their designee, the CRO, will assign site monitors to conduct regular site visits to the investigational facilities for the purpose of monitoring various aspects of the study. The Investigator must agree to allow personnel authorized by the Sponsor or the CRO direct access to the clinical (or associated) files and clinical study supplies (dispensing and storage areas) for all study subjects considered for study entry for the purpose of verifying entries made in the eCRF, and assist with their activities, if requested. Adequate time and space for monitoring visits should be made available by the Investigator.

The site must complete the eCRFs in a timely manner and on an ongoing basis to allow regular review by the study monitor.

Whenever a subject name is revealed on a document that is to be collected for the Sponsor, the name must be blacked out permanently by the site personnel, leaving the initials visible (or other appropriate de-identifying information), and annotated with the subject number as identification.

### 14 AMENDMENTS

Protocol modifications, except those intended to reduce immediate risk to study subjects, may be made only by the Sponsor. A protocol change intended to eliminate an apparent immediate hazard to subjects may be implemented immediately, provided the IRB/IEC is notified within 5 days.

Any permanent, significant change to the protocol must be handled as a protocol amendment. The written amendment must be submitted to the IRB/IEC and the Investigator must await approval before implementing the changes. The Sponsor will submit protocol amendments to the appropriate regulatory authorities for approval.

If, in the judgment of the IRB/IEC, the Investigator, and/or the Sponsor, the amendment to the protocol substantially changes the study design and/or increases the potential risk to the subject and/or has an impact on the subject's involvement as a study subject, the currently approved written ICF will require similar modification. In such cases, subjects will be required for to sign the amended informed consent prior to continued participation in the study.

# 15 STUDY REPORT AND PUBLICATIONS

The Sponsor or its designee is responsible for preparing and providing the appropriate regulatory authorities with clinical study reports according to the applicable regulatory requirements.

The publication policy of the Sponsor is discussed in the Investigator's Clinical Research Agreement.

# 16 STUDY DISCONTINUATION

Both the Sponsor and the Investigator reserve the right to terminate the study at the Investigator's site at any time. Should this be necessary, the Sponsor or a specified designee will inform the appropriate regulatory authorities of the termination of the study and the reasons for its termination, and the Investigator will inform the IRB/IEC of the same. In terminating the study, the Sponsor and the Investigator will assure that adequate consideration is given to the protection of the subjects' interests.

# 17 CONFIDENTIALITY

All information generated in this study is considered highly confidential and must not be disclosed to any person or entity not directly involved with the study unless prior written consent is gained from the Sponsor. However, authorized regulatory officials, IRB/IEC personnel, and the Sponsor and the Sponsor's authorized representatives are allowed full access to the records.

Identification of subjects and eCRFs shall be by initials (except in the United Kingdom) and screening and randomization numbers only. If required, the subject's full name may be made known to an authorized regulatory agency or other authorized official.
#### 18 REFERENCES

Belloni L, Li L, Palumbo GA, et al. HAPs hepatitis B virus (HBV) capsid inhibitors block core protein interaction with the viral minichromosome and host cell genes and affect cccDNA transcription and stability. Hepatology. 2013;58(4 suppl 1):277A.

Boyd, A, Lacombe, K, Lavocat, et al. Decay of ccc-DNA is slow and marks persistence of intrahepatic viral DNA synthesis under tenofovir in HIV-HBV co-infected patients. J Hepatol. 2016; 65:683–691.

European Association for the Study of the Liver (EASL) Clinical Practice Guidelines: Management of chronic hepatitis B virus infection. J Hepatol. 2012;57:167-185. European Medicines Agency. Guideline on Strategies to Identify and Mitigate Risks for First-In-Human Clinical Trials with Investigational Medicinal Products. London; 19 July 2007.

Gane EJ, Stedman CA, Hyland RH, et al. Nucleotide Polymerase Inhibitor Sofosbuvir plus Ribavirin for Hepatitis C. N Engl J Med 2013;368:34–44.

Gruffaz M et al. The nuclear function of hepatitis B capsid (HBc) protein is to inhibit IFN response very early after infection of hepatocytes. American Association for the Study of Liver Diseases (AASLD), The Liver Meeting 2013, November 01 - 05, 2013; Washington, DC. Abstract #136.

Guettouche T, Hnatyszyn HJ. Chronic hepatitis B and viral genotype: the clinical significance of determining HBV genotypes. Antivir Ther. 2005;10(5):593–604.

Heimbach JK, Kulik LM, Finn RS, et al. AASLD Guidelines for the Treatment of Hepatocellular Carcinoma. Hepatology. 2018;67(1):358–380.

Levey AS1, Stevens LA, et al. A new equation to estimate glomerular filtration rate. Ann Intern Med. 2009 May 5;150(9):604–612.

Liaw YF1, Leung N, Kao JH, et al. Asian-Pacific consensus statement on the management of chronic hepatitis B: a 2008 update. Hepatol Int. 2008 Sep;2(3):263–283.

Marcellin, P, Buti, M, et al. Kinetics of hepatitis B surface antigen loss in patients with HBeAg-positive chronic hepatitis B treated with tenofovir disoproxil fumarate. J Hepatology. 2014;61(6):1228–1237.

Ott JJ, Stevens GA, Groeger J, Wiersma ST. Global epidemiology of hepatitis B virus infection: New estimates of age-specific HBsAg seroprevalence and endemicity. Vaccine. 2012;30:2212–2219.

Seeger C, Zoulim F and Mason W, Hepadnaviruses, in Knipe DM and Howley PM eds. Fields Virology, 6th edition, Volume 2, chapter 68, 2013, Lippincott Williams & Wilkins, Philadelphia.

Stanaway JD, Flaxman AD, et al. The global burden of viral hepatitis from 1990 to 2013. Lancet. 2016 Sep 10;388(10049):1081–1088.

Wang Q, Luan W, Warren L, et al. Serum hepatitis B surface antigen correlates with tissue covalently closed circular DNA in patients with hepatitis B-associated hepatocellular carcinoma. J Med Virol. 2016 Feb;88(2):244–251.

World Health Organization. Hepatitis B: fact sheet. Updated July 2015. http://www.who.int/mediacentre/factsheets/fs204/en/. Accessed 22 March 2018.

# 19 APPENDICES

# 19.1 APPENDIX I – Names of Study Personnel

| Sponsor: | Assembly Biosciences |
|----------------------------------|-----------------------|
| Medical Monitor: | |
| Clinical Research Organizations: | PRA Health Sciences |
| | 4130 Parklake Avenue |
| | Raleigh, NC 27612 USA |

#### 19.2 APPENDIX II – Adverse Event Intensity Grading

TOXICITY GRADING OF LABORATORY ABNORMALITIES AND CLINICAL ADVERSE EVENTS. PUBLISH DATE: JULY 2017

Adapted from the U.S. National Institutes of Health (Division of AIDS) Table for Grading Severity of Adult Adverse Experiences (July 2017). Parameters within the table that have been modified for this study are designated by an asterisk (\*).

#### **MAJOR CLINICAL CONDITIONS**

#### Cardiovascular

| Parameter | Grade 1 Mild | Grade 2 Moderate | Grade 3 Severe | Grade 4 Potentially<br>Life- Threatening |
|---|---|---|---|---|
| Arrhythmia (by ECG or physical examination) Specify type, if applicable | No symptoms <u>AND</u> No intervention indicated | No symptoms <u>AND</u><br>Non-urgent<br>intervention indicated | Non-life-threatening<br>symptoms AND<br>Non-urgent<br>intervention<br>indicated | Life-threatening arrhythmia OR Urgent intervention indicated |
| Blood Pressure<br>Abnormalities | | | | |
| Hypertension (with the lowest reading taken after repeat testing during a visit) | 140 to < 160 mmHg<br>systolic<br>OR<br>90 to < 100 mmHg<br>diastolic | ≥ 160 to < 180<br>mmHg systolic<br><u>OR</u><br>≥ 100 to < 110 mmHg<br>diastolic | ≥ 180 mmHg systolic OR ≥ 110 mmHg diastolic | Life-threatening consequences in a participant not previously diagnosed with hypertension (e.g., malignant hypertension) OR Hospitalization indicated |
| Hypotension | No symptoms | Symptoms corrected<br>with oral fluid<br>replacement | Symptoms <u>AND</u> IV fluids indicated | Shock requiring use of vasopressors or mechanical assistance to maintain blood pressure |
| Cardiac Ischemia or<br>Infarction<br>Report only one | NA | NA | New symptoms with ischemia (stable angina) OR New testing consistent with ischemia | Unstable angina OR Acute myocardial infarction |
| Heart Failure | No symptoms <u>AND</u><br>Laboratory or cardiac<br>imaging abnormalities | Symptoms with mild to moderate activity or exertion | Symptoms at rest or with minimal activity or exertion (e.g., hypoxemia) OR Intervention indicated (e.g., oxygen) | Life-threatening consequences <u>OR</u> Urgent intervention indicated (e.g., vasoactive medications, ventricular assist device, heart transplant) |
| Hemorrhage<br>(with significant acute<br>blood loss) | NA | Symptoms <u>AND</u> No transfusion indicated | Symptoms <u>AND</u><br>Transfusion of ≤ 2 units<br>packed RBCs indicated | Life-threatening<br>hypotension <u>OR</u><br>Transfusion of > 2 units<br>packed RBCs indicated |

# Cardiovascular

| Parameter | Grade 1 Mild | Grade 2 Moderate | Grade 3 Severe | Grade 4 Potentially<br>Life- Threatening |
|---|---|---|---|---|
| Prolonged QTc<br>Interval <sup>1</sup> | 0.45 to 0.47 seconds | > 0.47 to 0.50 seconds | > 0.50 seconds <u>OR</u><br>≥ 0.06 seconds above<br>baseline | Life-threatening consequences (e.g., Torsade de pointes, other associated serious ventricular dysrhythmia) |
| Thrombosis<br>or Embolism<br>Report only one | NA | Symptoms <u>AND</u> No intervention indicated | Symptoms <u>AND</u><br>Intervention indicated | Life-threatening<br>embolic event (e.g.,<br>pulmonary embolism,<br>thrombus) |

<sup>1</sup> As per Bazett's formula.

Dermatologic

| Dermatologic | | | | Grade 4 Potentially |
|---|---|---|---|---|
| Parameter | Grade 1 Mild | Grade 2 Moderate | Grade 3 Severe | Life- Threatening |
| Alopecia (scalp only) | Detectable by study participant, caregiver, or physician AND Causing no or minimal interference with usual social & functional activities | Obvious on visual inspection AND Causing greater than minimal interference with usual social & functional activities | NA | NA |
| Bruising | Localized to one area | Localized to more than one area | Generalized | NA |
| Cellulitis | NA | Non-parenteral<br>treatment indicated<br>(e.g., oral antibiotics,<br>antifungals, antivirals) | IV treatment indicated (e.g., IV antibiotics, antifungals, antivirals) | Life-threatening consequences (e.g., sepsis, tissue necrosis) |
| Hyperpigmentation | Slight or localized causing no or minimal interference with usual social & functional activities | Marked or generalized causing greater than minimal interference with usual social & functional activities | NA | NA |
| Hypopigmentation | Slight or localized causing no or minimal interference with usual social & functional activities | Marked or generalized causing greater than minimal interference with usual social & functional activities | NA | NA |
| Petechiae | Localized to one area | Localized to more than one area | Generalized | NA |
| Pruritus <sup>3</sup> (without skin lesions) | Itching causing no or<br>minimal interference<br>with usual social &<br>functional activities | Itching causing greater<br>than minimal<br>interference with usual<br>social & functional<br>activities | Itching causing inability to perform usual social & functional activities | NA |
| Rash Specify type, if applicable | Localized rash | Diffuse rash <u>OR</u> Target lesions | Diffuse rash <u>AND</u> Vesicles or limited number of bullae or superficial ulcerations of mucous membrane limited to one site | Extensive or generalized bullous lesions <b>OR</b> Ulceration of mucous membrane involving 2 or more distinct mucosal sites OR Stevens-Johnson syndrome <b>OR</b> Toxic epidermal necrolysis |

<sup>3</sup> For pruritus associated with injections or infusions, see the Site Reactions to Injections and Infusions section.

## **Endocrine and Metabolic**

| Parameter | Grade 1 Mild | Grade 2 Moderate | Grade 3 Severe | Grade 4 Potentially Life-<br>Threatening |
|---|---|---|---|---|
| Diabetes Mellitus | Controlled without medication | Controlled with medication OR Modification of current medication regimen | Uncontrolled despite treatment modification OR Hospitalization for immediate glucose control indicated | Life-threatening consequences (e.g., ketoacidosis, hyperosmolar non- ketotic coma, end organ failure) |
| Gynecomastia | Detectable by study participant, caregiver, or physician AND Causing no or minimal interference with usual social & functional activities | Obvious on visual inspection AND Causing pain with greater than minimal interference with usual social & functional activities | Disfiguring changes <u>AND</u> Symptoms requiring intervention or causing inability to perform usual social & functional activities | NA |
| Hyperthyroidism | No symptoms <u>AND</u><br>Abnormal laboratory<br>value | Symptoms causing greater than minimal interference with usual social & functional activities <u>OR</u> Thyroid suppression therapy indicated | Symptoms causing inability to perform usual social & functional activities OR Uncontrolled despite treatment modification | Life-threatening consequences (e.g., thyroid storm) |
| Hypothyroidism | No symptoms <u>AND</u><br>Abnormal laboratory<br>value | Symptoms causing greater than minimal interference with usual social & functional activities <u>OR</u> Thyroid replacement therapy indicated | Symptoms causing inability to perform usual social & functional activities OR Uncontrolled despite treatment modification | Life-threatening consequences (e.g., myxedema coma) |
| Lipoatrophy <sup>4</sup> | Detectable by study participant, caregiver, or physician AND Causing no or minimal interference with usual social & functional activities | Obvious on visual inspection AND Causing greater than minimal interference with usual social & functional activities | Disfiguring changes | NA |
| Lipohypertrophy <sup>5</sup> | Detectable by study participant, caregiver, or physician AND Causing no or minimal interference with usual social & functional activities | Obvious on visual inspection AND Causing greater than minimal interference with usual social & functional activities | Disfiguring changes | NA |

<sup>4</sup> Definition: A disorder characterized by fat loss in the face, extremities, and buttocks.

<sup>5</sup> Definition: A disorder characterized by abnormal fat accumulation on the back of the neck, breasts, and abdomen.

## Gastrointestinal

| Parameter | Grade 1 Mild | Grade 2 Moderate | Grade 3 Severe | Grade 4 Potentially<br>Life- Threatening |
|---|---|---|---|---|
| Anorexia | Loss of appetite without decreased oral intake | Loss of appetite<br>associated with decreased<br>oral intake without<br>significant weight loss | Loss of appetite<br>associated with<br>significant weight loss | Life-threatening consequences OR Aggressive intervention indicated (e.g., tube feeding, total parenteral nutrition) |
| Ascites | No symptoms | Symptoms AND Intervention indicated (e.g., diuretics, therapeutic paracentesis) | Symptoms recur or persist despite intervention | Life-threatening consequences |
| Bloating or Distension<br>Report only one | Symptoms causing no or minimal interference with usual social & functional activities | Symptoms causing greater than minimal interference with usual social & functional activities | Symptoms causing inability to perform usual social & functional activities | NA |
| Cholecystitis | NA | Symptoms AND Medical intervention indicated | Radiologic, endoscopic, or operative intervention indicated | Life-threatening consequences (e.g., sepsis, perforation) |
| Constipation | NA | Persistent constipation<br>requiring regular use of<br>dietary modifications,<br>laxatives, or enemas | Obstipation with manual evacuation indicated | Life-threatening consequences (e.g., obstruction) |
| Diarrhea | Transient or intermittent episodes of unformed stools OR Increase of ≤3 stools over baseline per 24-hour period | Persistent episodes of<br>unformed to watery<br>stools OR Increase of 4 to<br>6 stools over baseline per<br>24-hour period | Increase of ≥7 stools per<br>24-hour period OR IV<br>fluid replacement<br>indicated | Life-threatening<br>consequences (e.g.,<br>hypotensive shock) |
| Dysphagia or Odynophagia Report only one and specify location | Symptoms but able to eat usual diet | Symptoms causing<br>altered dietary intake<br>with no intervention<br>indicated | Symptoms causing severely altered dietary intake with intervention indicated | Life-threatening reduction in oral intake |

## Gastrointestinal

| Parameter | Grade 1 Mild | Grade 2 Moderate | Grade 3 Severe | Grade 4 Potentially<br>Life- Threatening |
|---|---|---|---|---|
| Gastrointestinal<br>Bleeding | Not requiring intervention other than iron supplement | Endoscopic intervention indicated | Transfusion indicated | Life-threatening consequences (e.g., hypotensive shock) |
| Mucositis or Stomatitis Report only one and specify location | Mucosal erythema | Patchy pseudomembranes or ulcerations | Confluent<br>pseudomembranes or<br>ulcerations OR Mucosal<br>bleeding with minor<br>trauma | Life-threatening consequences (e.g., aspiration, choking) OR Tissue necrosis OR Diffuse spontaneous mucosal bleeding |
| Nausea | Transient (<24 hours)<br>or intermittent AND<br>No or minimal<br>interference with oral<br>intake | Persistent nausea<br>resulting in decreased<br>oral intake for 24 to 48<br>hours | Persistent nausea<br>resulting in minimal oral<br>intake for >48 hours OR<br>Rehydration indicated<br>(e.g., IV fluids) | Life-threatening<br>consequences (e.g.,<br>hypotensive shock) |
| Pancreatitis | NA | Symptoms with hospitalization not indicated | Symptoms with hospitalization indicated | Life-threatening<br>consequences (e.g.,<br>circulatory failure,<br>hemorrhage, sepsis) |
| Perforation (colon or rectum) | NA | NA | Intervention indicated | Life-threatening consequences |
| Proctitis | Rectal discomfort with no intervention indicated | Symptoms causing greater than minimal interference with usual social & functional activities OR Medical intervention indicated | Symptoms causing inability to perform usual social & functional activities OR Operative intervention indicated | Life-threatening consequences (e.g., perforation) |
| Rectal Discharge | Visible discharge | Discharge requiring the use of pads | NA | NA |
| Vomiting | Transient or intermittent AND No or minimal interference with oral intake | Frequent episodes with no or mild dehydration | Persistent vomiting resulting in orthostatic hypotension OR Aggressive rehydration indicated (e.g., IV fluids) | Life-threatening<br>consequences (e.g.,<br>hypotensive shock) |

## Musculoskeletal

| Parameter | Grade 1 Mild | Grade 2 Moderate | Grade 3 Severe | Grade 4 Potentially<br>Life- Threatening |
|---|---|---|---|---|
| Arthralgia | Joint pain causing no or minimal interference with usual social & functional activities | Joint pain causing greater than minimal interference with usual social & functional activities | Joint pain causing inability to perform usual social & functional activities | Disabling joint pain<br>causing inability to<br>perform basic self-care<br>functions |
| Arthritis | Stiffness or joint<br>swelling causing no or<br>minimal interference<br>with usual social &<br>functional activities | Stiffness or joint<br>swelling causing greater<br>than minimal<br>interference with usual<br>social & functional<br>activities | Stiffness or joint<br>swelling causing<br>inability to perform<br>usual social &<br>functional activities | Disabling joint stiffness<br>or swelling causing<br>inability to perform<br>basic self-care functions |
| Myalgia (generalized) | Muscle pain causing no or minimal interference with usual social & functional activities | Muscle pain causing greater than minimal interference with usual social & functional activities | Muscle pain causing inability to perform usual social & functional activities | Disabling muscle pain<br>causing inability to<br>perform basic self-care<br>functions |
| Osteonecrosis | NA | No symptoms but with<br>radiographic findings<br>AND No operative<br>intervention indicated | Bone pain with radiographic findings OR Operative intervention indicated | Disabling bone pain<br>with radiographic<br>findings causing<br>inability to perform<br>basic self-care functions |
| Osteopenia <sup>6</sup> | | | | |
| ≥30 years of age | BMD t-score -2.5 to -1 | NA | NA | NA |
| <30 years of age | BMD z-score -2 to -1 | NA | NA | NA |
| Osteoporosis <sup>6</sup><br>≥30 years of age | NA | BMD t-score <-2.5 | Pathologic fracture<br>(e.g., compression<br>fracture causing loss of<br>vertebral height) | Pathologic fracture causing life-threatening consequences |
| <30 years of age | NA | BMD z-score <-2 | Pathologic fracture<br>(e.g., compression<br>fracture causing loss of<br>vertebral height) | Pathologic fracture causing life-threatening consequences |

6 BMD t and z scores can be found in: Kanis JA on behalf of the WHO Scientific Group (2007). Assessment of osteoporosis at the primary health-care level. Technical Report. WHO Collaborating Centre for Metabolic Bone Diseases, University of Sheffield, UK. 2007: Printed by the University of Sheffield.

| T A | | | | • |
|-----|-----|----|---|-----|
| | AII | MA | | gic |
| 1.4 | Cu | ıv | ш | ยเ |

| Neurologic | 1 | T | 1 | T |
|---|---|---|---|---|
| Parameter | Grade 1 Mild | Grade 2 Moderate | Grade 3 Severe | Grade 4 Potentially Life- Threatening |
| Acute CNS Ischemia | NA | NA | Transient ischemic attack | Cerebral vascular<br>accident (e.g., stroke<br>with neurological<br>deficit) |
| Altered Mental Status (for Dementia, see Cognitive, Behavioral, or Attentional Disturbance below) | Changes causing no or minimal interference with usual social & functional activities | Mild lethargy or<br>somnolence causing<br>greater than minimal<br>interference with usual<br>social & functional<br>activities | Confusion, memory impairment, lethargy, or somnolence causing inability to perform usual social & functional activities | Delirium OR<br>Obtundation OR Coma |
| Ataxia | Symptoms causing no or minimal interference with usual social & functional activities OR No symptoms with ataxia detected on examination | Symptoms causing greater than minimal interference with usual social & functional activities | Symptoms causing inability to perform usual social & functional activities | Disabling symptoms causing inability to perform basic self-care functions |
| Cognitive, Behavioral, or Attentional Disturbance (includes dementia and attention deficit disorder) Specify type, if applicable | Disability causing no or minimal interference with usual social & functional activities OR Specialized resources not indicated | Disability causing greater than minimal interference with usual social & functional activities OR Specialized resources on part- time basis indicated | Disability causing inability to perform usual social & functional activities OR Specialized resources on a full-time basis indicated | Disability causing inability to perform basic self-care functions OR Institutionalization indicated |
| Headache | Symptoms causing no or minimal interference with usual social & functional activities | Symptoms causing greater than minimal interference with usual social & functional activities | Symptoms causing inability to perform usual social & functional activities | Symptoms causing inability to perform basic self-care functions OR Hospitalization indicated OR Headache with significant impairment of alertness or other neurologic function |
| Neuromuscular<br>Weakness (includes<br>myopathy and<br>neuropathy) Specify<br>type, if applicable | Minimal muscle weakness causing no or minimal interference with usual social & functional activities OR No symptoms with decreased strength on examination | Muscle weakness causing greater than minimal interference with usual social & functional activities | Muscle weakness causing inability to perform usual social & functional activities | Disabling muscle weakness causing inability to perform basic self-care functions OR Respiratory muscle weakness impairing ventilation |
| Neurosensory Alteration (includes paresthesia and painful neuropathy) Specify type, if applicable | Minimal paresthesia causing no or minimal interference with usual social & functional activities OR No symptoms with sensory alteration on examination | Sensory alteration or<br>paresthesia causing<br>greater than minimal<br>interference with usual<br>social & functional<br>activities | Sensory alteration or<br>paresthesia causing<br>inability to perform<br>usual social &<br>functional activities | Disabling sensory<br>alteration or paresthesia<br>causing inability to<br>perform basic self-care<br>functions |

Neurologic

| Parameter | Grade 1 Mild | Grade 2 Moderate | Grade 3 Severe | Grade 4 Potentially<br>Life- Threatening |
|---|---|---|---|---|
| Seizures<br>New Onset Seizure | NA | NA | 1 to 3 seizures | Prolonged and<br>repetitive seizures (e.g.,<br>status epilepticus) OR<br>Difficult to control (e.g.,<br>refractory epilepsy) |
| Pre-existing Seizure | NA | Increased frequency<br>from previous level of<br>control without change<br>in seizure character | Change in seizure character either in duration or quality (e.g., severity or focality) | Prolonged and repetitive<br>seizures (e.g., status<br>epilepticus) OR Difficult<br>to control (e.g.,<br>refractory epilepsy) |
| Syncope | Near syncope without loss of consciousness (e.g., presyncope) | Loss of consciousness with no intervention indicated | Loss of consciousness<br>AND Hospitalization or<br>intervention required | NA |

Pregnancy, Puerperium, and Perinatal

| Parameter | Grade 1 Mild | Grade 2 Moderate | Grade 3 Severe | Grade 4 Potentially<br>Life- Threatening |
|---|---|---|---|---|
| Stillbirth (report using mother's participant ID) Report only one | NA | NA | Fetal death occurring at ≥20 weeks gestation | NA |
| Preterm Birth (report using mother's participant ID) | Live birth at 34 to <37 weeks gestational age | Live birth at 28 to <34 weeks gestational age | Live birth at 24 to <28 weeks gestational age | Live birth at <24 weeks gestational age |
| Spontaneous Abortion<br>or Miscarriage <sup>7</sup> (report<br>using mother's<br>participant ID) | Chemical pregnancy | Uncomplicated spontaneous abortion or miscarriage | Complicated spontaneous abortion or miscarriage | NA |
| Report only one | | | | |

<sup>7</sup> Definition: A pregnancy loss occurring at <20 weeks gestational age.

# Psychiatric

| Parameter | Grade 1 Mild | Grade 2 Moderate | Grade 3 Severe | Grade 4 Potentially<br>Life- Threatening |
|---|---|---|---|---|
| Insomnia | Mild difficulty falling<br>asleep, staying asleep,<br>or waking up early<br>causing no or minimal<br>interference with usual<br>social & functional<br>activities | Moderate difficulty falling asleep, staying asleep, or waking up early causing more than minimal interference with usual social & functional activities | Severe difficulty falling asleep, staying asleep, or waking up early causing inability to perform usual social & functional activities requiring intervention or hospitalization | NA |
| Psychiatric Disorders<br>(includes anxiety,<br>depression, mania, and<br>psychosis)<br>Specify disorder | Symptoms with intervention not indicated OR Behavior causing no or minimal interference with usual social & functional activities | Symptoms with intervention indicated OR Behavior causing greater than minimal interference with usual social & functional activities | Symptoms with hospitalization indicated OR Behavior causing inability to perform usual social & functional activities | Threatens harm to self<br>or others OR Acute<br>psychosis OR Behavior<br>causing inability to<br>perform basic self-care<br>functions |
| Suicidal Ideation or<br>Attempt<br>Report only one | Preoccupied with<br>thoughts of death AND<br>No wish to kill oneself | Preoccupied with<br>thoughts of death AND<br>Wish to kill oneself<br>with no specific plan or<br>intent | Thoughts of killing<br>oneself with partial or<br>complete plans but no<br>attempt to do so OR<br>Hospitalization<br>indicated | Suicide attempted |

Respiratory

| Parameter | Grade 1 Mild | Grade 2 Moderate | Grade 3 Severe | Grade 4 Potentially<br>Life- Threatening |
|---|---|---|---|---|
| Acute Bronchospasm | Forced expiratory volume in 1 second or peak flow reduced to ≥70 to <80% OR Mild symptoms with intervention not indicated | Forced expiratory volume in 1 second or peak flow 50 to <70% OR Symptoms with intervention indicated OR Symptoms causing greater than minimal interference with usual social & functional activities | Forced expiratory volume in 1 second or peak flow 25 to <50% OR Symptoms causing inability to perform usual social & functional activities | Forced expiratory<br>volume in 1 second or<br>peak flow <25% OR<br>Life-threatening<br>respiratory or<br>hemodynamic<br>compromise OR<br>Intubation |
| Dyspnea or<br>Respiratory Distress<br>Report only one | Dyspnea on exertion with no or minimal interference with usual social & functional activities OR Wheezing OR Minimal increase in respiratory rate for age | Dyspnea on exertion causing greater than minimal interference with usual social & functional activities OR Nasal flaring OR Intercostal retractions OR Pulse oximetry 90 to <95% | Dyspnea at rest causing inability to perform usual social & functional activities OR Pulse oximetry <90% | Respiratory failure with<br>ventilator support<br>indicated (e.g., CPAP,<br>BPAP, intubation) |

## Sensory

| Parameter | Grade 1 Mild | Grade 2 Moderate | Grade 3 Severe | Grade 4 Potentially<br>Life- Threatening |
|---|---|---|---|---|
| Hearing Loss | NA | Hearing aid or intervention not indicated | Hearing aid or intervention indicated | Profound bilateral<br>hearing loss (>80 dB at<br>2 kHz and above) OR<br>Non-serviceable hearing<br>(i.e., >50 dB audiogram<br>and <50% speech<br>discrimination) |
| Tinnitus | Symptoms causing no or minimal interference with usual social & functional activities with intervention not indicated | Symptoms causing greater than minimal interference with usual social & functional activities with intervention indicated | Symptoms causing inability to perform usual social & functional activities | NA |
| Uveitis | No symptoms AND Detectable on examination | Anterior uveitis with symptoms OR Medical intervention indicated | Posterior or pan-uveitis<br>OR Operative<br>intervention indicated | Disabling visual loss in affected eye(s) |
| Vertigo | Vertigo causing no or<br>minimal interference<br>with usual social &<br>functional activities | Vertigo causing greater<br>than minimal<br>interference with usual<br>social & functional<br>activities | Vertigo causing inability to perform usual social & functional activities | Disabling vertigo<br>causing inability to<br>perform basic self-care<br>functions |
| Visual Changes<br>(assessed from<br>baseline) | Visual changes causing no or minimal interference with usual social & functional activities | Visual changes causing greater than minimal interference with usual social & functional activities | Visual changes causing inability to perform usual social & functional activities | Disabling visual loss in affected eye(s) |

#### **Systemic**

| Systemic | | | | |
|---|---|---|---|---|
| Parameter | Grade 1 Mild | Grade 2 Moderate | Grade 3 Severe | Grade 4 Potentially Life- Threatening |
| Acute Allergic<br>Reaction | Localized urticaria<br>(wheals) with no<br>medical intervention<br>indicated | Localized urticaria with intervention indicated OR Mild angioedema with no intervention indicated | Generalized urticaria OR Angioedema with intervention indicated OR Symptoms of mild bronchospasm | Acute anaphylaxis OR<br>Life-threatening<br>bronchospasm OR<br>Laryngeal edema |
| Chills | Symptoms causing no or minimal interference with usual social & functional activities | Symptoms causing greater than minimal interference with usual social & functional activities | Symptoms causing inability to perform usual social & functional activities | NA |
| Cytokine Release<br>Syndrome <sup>8</sup> | Mild signs and<br>symptoms AND<br>Therapy (i.e., antibody<br>infusion) interruption<br>not indicated | Therapy (i.e., antibody infusion) interruption indicated AND Responds promptly to symptomatic treatment OR Prophylactic medications indicated for ≤24 hours | Prolonged severe signs<br>and symptoms OR<br>Recurrence of<br>symptoms following<br>initial improvement | Life-threatening<br>consequences (e.g.,<br>requiring pressor or<br>ventilator support) |
| Fatigue or Malaise<br>Report only one | Symptoms causing no or minimal interference with usual social & functional activities | Symptoms causing greater than minimal interference with usual social & functional activities | Symptoms causing inability to perform usual social & functional activities | Incapacitating<br>symptoms of fatigue or<br>malaise causing<br>inability to perform<br>basic self-care functions |
| Fever (non-axillary temperatures only) | 38.0 to <38.6°C or<br>100.4 to <101.5°F | ≥38.6 to <39.3°C or<br>≥101.5 to <102.7°F | ≥39.3 to <40.0°C or<br>≥102.7 to <104.0°F | ≥40.0°C or<br>≥104.0°F |
| Pain 9 (not associated with study agent injections and not specified elsewhere) Specify location | Pain causing no or<br>minimal interference<br>with usual social &<br>functional activities | Pain causing greater<br>than minimal<br>interference with usual<br>social & functional<br>activities | Pain causing inability to perform usual social & functional activities | Disabling pain causing inability to perform basic self-care functions OR Hospitalization indicated |
| Serum Sickness <sup>10</sup> | Mild signs and symptoms | Moderate signs and<br>symptoms AND<br>Intervention indicated<br>(e.g., antihistamines) | Severe signs and<br>symptoms AND Higher<br>level intervention<br>indicated (e.g., steroids<br>or IV fluids) | Life-threatening consequences (e.g., requiring pressor or ventilator support) |
| Underweight <sup>11</sup> | WHO BMI z-score<br><-1 to -2 | WHO BMI z-score<br><-2 to -3 | WHO BMI z-score <-3 | WHO BMI z-score <-3 with life-threatening consequences |
| Unintentional Weight<br>Loss<br>(excludes postpartum<br>weight loss) | NA | 5 to <9% loss in body<br>weight from baseline | ≥9 to <20% loss in body weight from baseline | ≥20% loss in body<br>weight from baseline<br>OR Aggressive<br>intervention indicated<br>(e.g., tube feeding, total<br>parenteral nutrition) |

<sup>8</sup> Definition: A disorder characterized by nausea, headache, tachycardia, hypotension, rash, and/or shortness of breath.

<sup>9</sup> For pain associated with injections or infusions, see the Site Reactions to Injections and Infusions section.

<sup>10</sup> Definition: A disorder characterized by fever, arthralgia, myalgia, skin eruptions, lymphadenopathy, marked discomfort, and/or dyspnea.

<sup>11</sup> WHO reference tables may be accessed by clicking the desired age range or by accessing the following URL: http://www.who.int/growthref/who2007\_bmi\_for\_age/en/ for participants >5 to 19 years of age

Urinary

| Parameter | Grade 1 Mild | Grade 2 Moderate | Grade 3 Severe | Grade 4 Potentially<br>Life- Threatening |
|---|---|---|---|---|
| Urinary Tract<br>Obstruction | NA | Signs or symptoms of urinary tract obstruction | Signs or symptoms of urinary tract obstruction | Obstruction causing life-threatening |
| | | without hydronephrosis or renal dysfunction | with hydronephrosis or renal dysfunction | consequences |

## Site Reactions to Injections and Infusions

| Parameter | Grade 1 Mild | Grade 2 Moderate | Grade 3 Severe | Grade 4 Potentially<br>Life- Threatening |
|---|---|---|---|---|
| Injection Site Pain or<br>Tenderness<br>Report only one | Pain or tenderness<br>causing no or minimal<br>limitation of use of limb | Pain or tenderness<br>causing greater than<br>minimal limitation of<br>use of limb | Pain or tenderness<br>causing inability to<br>perform usual social &<br>functional activities | Pain or tenderness<br>causing inability to<br>perform basic self-care<br>function OR<br>Hospitalization<br>indicated |
| Injection Site<br>Erythema or Redness<br>12<br>Report only one | 2.5 to <5 cm in diameter OR 6.25 to <25 cm <sup>2</sup> surface area AND Symptoms causing no or minimal interference with usual social & functional activities | ≥5 to <10 cm in<br>diameter OR ≥25 to<br><100 cm² surface area<br>OR Symptoms causing<br>greater than minimal<br>interference with usual<br>social & functional<br>activities | ≥10 cm in diameter OR<br>≥100 cm² surface area<br>OR Ulceration OR<br>Secondary infection OR<br>Phlebitis OR Sterile<br>abscess OR Drainage<br>OR Symptoms causing<br>inability to perform<br>usual social &<br>functional activities | Potentially life-<br>threatening<br>consequences (e.g.,<br>abscess, exfoliative<br>dermatitis, necrosis<br>involving dermis or<br>deeper tissue) |
| Injection Site<br>Induration or Swelling<br>Report only one | Same as for Injection Site Erythema or Redness, >15 years of age | Same as for Injection<br>Site Erythema or<br>Redness, >15 years of<br>age | Same as for Injection<br>Site Erythema or<br>Redness, >15 years of<br>age | Same as for Injection Site Erythema or Redness, >15 years of age |
| Injection Site Pruritus | Itching localized to the injection site that is relieved spontaneously or in <48 hours of treatment | Itching beyond the injection site that is not generalized OR Itching localized to the injection site requiring ≥48 hours treatment | Generalized itching causing inability to perform usual social & functional activities | NA |

<sup>12</sup> Injection Site Erythema or Redness should be evaluated and graded using the greatest single diameter or measured surface area.

**Laboratory Values\*: Chemistries** 

| Laboratory Value | s*: Chemistries | | | |
|---|---|---|---|---|
| Parameter | Grade 1 Mild | Grade 2 Moderate | Grade 3 Severe | Grade 4 Potentially<br>Life- Threatening |
| Acidosis | NA | pH≤7.3 to <lln< td=""><td>pH&lt;7.3 without life-<br/>threatening<br/>consequences</td><td>pH&lt;7.3 with life-<br/>threatening<br/>consequences</td></lln<> | pH<7.3 without life-<br>threatening<br>consequences | pH<7.3 with life-<br>threatening<br>consequences |
| Albumin, Low | 3.0 to < LLN | $\geq$ 2.0 to < 3.0 | < 2.0 | NA |
| (g/dL; g/L) | 30 to < LLN | $\geq 20$ to $< 30$ | < 20 | |
| Alkaline Phosphatase,<br>High | 1.25 to < 2.5 x ULN | 2.5 to < 5.0 x ULN | 5.0 to < 10.0 x ULN | ≥ 10.0 x ULN |
| Alkalosis | NA | pH > ULN to ≤ 7.5 | pH > 7.5 without life-<br>threatening<br>consequences | pH > 7.5 with life-<br>threatening<br>consequences |
| ALT or SGPT, High Report only one | 1.25 to < 2.5 x ULN | 2.5 to < 5.0 x ULN | 5.0 to < 10.0 x ULN | ≥ 10.0 x ULN |
| Amylase (Pancreatic) or Amylase (Total), High Report only one | 1.1 to <1.5×ULN | 1.5 to <3.0×ULN | 3.0 to <5.0×ULN | ≥5.0×ULN |
| AST or SGOT, High Report only one | 1.25 to < 2.5 x ULN | 2.5 to < 5.0 x ULN | 5.0 to < 10.0 x ULN | ≥ 10.0 x ULN |
| Bicarbonate, Low (mEq/L; mmol/L) | 16.0 to <lln 16.0="" <lln<="" td="" to=""><td>11.0 to &lt;16.0 <i>11.0 to</i> &lt;16.0</td><td>8.0 to &lt;11.0<br/>8.0 to &lt;11.0</td><td>&lt;8.0<br/>&lt;8.0</td></lln> | 11.0 to <16.0 <i>11.0 to</i> <16.0 | 8.0 to <11.0<br>8.0 to <11.0 | <8.0<br><8.0 |
| Bilirubin Direct Bilirubin, High | NA | NA | > ULN with other signs<br>and symptoms of<br>hepatotoxicity. | > ULN with life-<br>threatening<br>consequences (e.g.,<br>signs and symptoms of<br>liver failure) |
| Total Bilirubin, High | 1.1 to <1.6×ULN | 1.6 to <2.6×ULN | 2.6 to <5.0×ULN | ≥5.0×ULN |
| Calcium, High (mg/dL; mmol/L) | 10.6 to <11.5<br>2.65 to <2.88 | 11.5 to <12.5<br>2.88 to <3.13 | 12.5 to <13.5<br>3.13 to <3.38 | ≥3.5<br>≥3.38 |
| Calcium (Ionized), High (mg/dL; mmol/L) | >ULN to <6.0<br>>ULN to <1.5 | 6.0 to <6.4<br>1.5 to <1.6 | 6.4 to <7.2<br>1.6 to <1.8 | ≥7.2<br>≥1.8 |
| Calcium, Low (mg/dL; mmol/L) | 7.8 to <8.4<br>1.95 to <2.10 | 7.0 to <7.8<br>1.75 to <1.95 | 6.1 to <7.0<br>1.53 to <1.75 | <6.1<br><1.53 |
| Calcium (Ionized),<br>Low (mg/dL; mmol/L) | <lln 4.0<br="" to=""><lln 1.0<="" td="" to=""><td>3.6 to &lt;4.0<br/>0.9 to &lt;1.0</td><td>3.2 to &lt;3.6<br/>0.8 to &lt;0.9</td><td>&lt;3.2<br/>&lt;0.8</td></lln></lln> | 3.6 to <4.0<br>0.9 to <1.0 | 3.2 to <3.6<br>0.8 to <0.9 | <3.2<br><0.8 |
| Cardiac Troponin I,<br>High | NA | NA | NA | Levels consistent with<br>myocardial infarction or<br>unstable angina as<br>defined by the local<br>laboratory |
| Creatine Kinase, High | 3 to <6×ULN | 6 to <10×ULN | 10 to <20×ULN | ≥20×ULN |
| Creatinine, High *Report only one | 1.1 to 1.3×ULN | >1.3 to 1.8×ULN OR<br>Increase to 1.3 to<br><1.5×participant's<br>baseline | >1.8 to <3.5×ULN OR<br>Increase to 1.5 to<br><2.0×participant's<br>baseline | ≥3.5×ULN OR Increase of ≥2.0×participant's baseline |
| Creatinine Clearance 13 or eGFR, Low *Report only one | NA | <90 to 60 ml/min or<br>ml/min/1.73 m <sup>2</sup> OR 10<br>to <30% decrease from<br>participant's baseline | <60 to 30 ml/min or<br>ml/min/1.73 m <sup>2</sup> OR 30<br>to <50% decrease from<br>participant's baseline | <30 ml/min or<br>ml/min/1.73 m² OR<br>≥50% decrease from<br>participant's baseline or<br>dialysis needed |

<sup>\*</sup>Reminder: Choose the method that selects for the higher grade.

# **Laboratory Values\*: Chemistries**

| Laboratory Values*: | Grade 1 Mild | Grade 2 Moderate | Grade 3 Severe | Grade 4 Potentially Life- Threatening |
|---|---|---|---|---|
| Acidosis | NA NA | pH≤7.3 to <lln< td=""><td>pH&lt;7.3 without life-<br/>threatening<br/>consequences</td><td>pH&lt;7.3 with life-<br/>threatening<br/>consequences</td></lln<> | pH<7.3 without life-<br>threatening<br>consequences | pH<7.3 with life-<br>threatening<br>consequences |
| Albumin, Low<br>(g/dL; g/L) | 3.0 to < LLN<br>30 to < LLN | $\geq 2.0 \text{ to} < 3.0$<br>$\geq 20 \text{ to} < 30$ | < 2.0<br>< 20 | NA |
| Alkaline Phosphatase, High | 1.25 to < 2.5 x<br>ULN | 2.5 to < 5.0 x ULN | 5.0 to < 10.0 x ULN | ≥ 10.0 x ULN |
| Alkalosis | NA | pH > ULN to ≤ 7.5 | pH > 7.5 without life-<br>threatening<br>consequences | pH > 7.5 with life-<br>threatening<br>consequences |
| ALT or SGPT, High Report only one | 1.25 to < 2.5 x<br>ULN | 2.5 to < 5.0 x ULN | 5.0 to < 10.0 x ULN | ≥ 10.0 x ULN |
| Amylase (Pancreatic) or<br>Amylase (Total), High<br>Report only one | 1.1 to <1.5×ULN | 1.5 to <3.0×ULN | 3.0 to <5.0×ULN | ≥5.0×ULN |
| AST or SGOT, High Report only one | 1.25 to < 2.5 x<br>ULN | 2.5 to < 5.0 x ULN | 5.0 to < 10.0 x ULN | ≥ 10.0 x ULN |
| Bicarbonate, Low (mEq/L; mmol/L) | 16.0 to <lln<br>16.0 to <lln< td=""><td>11.0 to &lt;16.0 <i>11.0 to</i> &lt;16.0</td><td>8.0 to &lt;11.0<br/>8.0 to &lt;11.0</td><td>&lt;8.0<br/>&lt;8.0</td></lln<></lln<br> | 11.0 to <16.0 <i>11.0 to</i> <16.0 | 8.0 to <11.0<br>8.0 to <11.0 | <8.0<br><8.0 |
| Bilirubin Direct Bilirubin, High | NA | NA | > ULN with other signs<br>and symptoms of<br>hepatotoxicity. | > ULN with life-<br>threatening<br>consequences (e.g., signs<br>and symptoms of liver<br>failure) |
| Total Bilirubin, High | 1.1 to <1.6×ULN | 1.6 to <2.6×ULN | 2.6 to <5.0×ULN | ≥5.0×ULN |
| Calcium, High (mg/dL; mmol/L) | 10.6 to <11.5<br>2.65 to <2.88 | 11.5 to <12.5<br>2.88 to <3.13 | 12.5 to <13.5<br>3.13 to <3.38 | ≥3.5<br>≥3.38 |
| Calcium (Ionized), High (mg/dL; mmol/L) | >ULN to <6.0<br>>ULN to <1.5 | 6.0 to <6.4<br>1.5 to <1.6 | 6.4 to <7.2<br>1.6 to <1.8 | ≥7.2<br>≥1.8 |
| Calcium, Low (mg/dL; mmol/L) | 7.8 to <8.4<br>1.95 to <2.10 | 7.0 to <7.8<br>1.75 to <1.95 | 6.1 to <7.0<br>1.53 to <1.75 | <6.1<br><1.53 |
| Calcium (Ionized), Low (mg/dL; mmol/L) | <lln 4.0<br="" to=""><lln 1.0<="" td="" to=""><td>3.6 to &lt;4.0<br/>0.9 to &lt;1.0</td><td>3.2 to &lt;3.6<br/>0.8 to &lt;0.9</td><td>&lt;3.2<br/>&lt;0.8</td></lln></lln> | 3.6 to <4.0<br>0.9 to <1.0 | 3.2 to <3.6<br>0.8 to <0.9 | <3.2<br><0.8 |
| Cardiac Troponin I, High | NA | NA | NA | Levels consistent with<br>myocardial infarction or<br>unstable angina as<br>defined by the local<br>laboratory |
| Creatine Kinase, High | 3 to <6×ULN | 6 to <10×ULN | 10 to <20×ULN | ≥20×ULN |
| Creatinine, High *Report only one | 1.1 to 1.3×ULN | >1.3 to 1.8×ULN OR<br>Increase to 1.3 to<br><1.5×participant's<br>baseline | >1.8 to <3.5×ULN OR<br>Increase to 1.5 to<br><2.0×participant's<br>baseline | ≥3.5×ULN OR Increase of ≥2.0×participant's baseline |
| Creatinine Clearance <sup>13</sup> or eGFR, Low *Report only one | NA | <90 to 60 ml/min or<br>ml/min/1.73 m <sup>2</sup> OR 10<br>to <30% decrease from<br>participant's baseline | <60 to 30 ml/min or<br>ml/min/1.73 m <sup>2</sup> OR 30<br>to <50% decrease from<br>participant's baseline | <30 ml/min or<br>ml/min/1.73 m² OR<br>≥50% decrease from<br>participant's baseline or<br>dialysis needed |

### **Laboratory Values\*: Chemistries**

| Laboratory values . ( | | | | Grade 4 Potentially |
|---|---|---|---|---|
| Parameter | Grade 1 Mild | Grade 2 Moderate | Grade 3 Severe | Life- Threatening |
| Glucose (mg/dL; mmol/L) Fasting, High | 110 to 125 | >125 to 250 | >250 to 500 | ≥500 |
| | 6.11 to <6.95 | 6.95 to <13.89 | 13.89 to <27.75 | ≥27.75 |
| Nonfasting, High | 116 to 160 | >160 to 250 | >250 to 500 | ≥500 |
| | 6.44 to <8.89 | 8.89 to <13.89 | 13.89 to <27.75 | ≥27.75 |
| Glucose, Low (mg/dL; mmol/L) | 55 to 64 | 40 to <55 | 30 to <40 | <30 |
| | 3.05 to <3.55 | 2.22 to <3.05 | 1.67 to <2.22 | <1.67 |
| Lactate, High | ULN to<br><2.0×ULN<br>without acidosis | ≥2.0×ULN without acidosis | Increased lactate with pH <7.3 without life-threatening consequences | Increased lactate with pH <7.3 with life-threatening consequences |
| Lipase, High | 1.1 to <1.5×ULN | 1.5 to <3.0×ULN | 3.0 to <5.0×ULN | ≥5.0×ULN |
| <b>Lipid Disorders</b> (mg/dL; mmol/L) | 200 to <240 | 240 to <300 | ≥300 | NA |
| Cholesterol, Fasting, High | 5.18 to <6.19 | 6.19 to <7.77 | ≥7.77 | |
| LDL, Fasting, High | 130 to <160<br>3.37 to <4.12 | 160 to <190<br>4.12 to <4.90 | ≥190<br>≥4.90 | NA |
| Triglycerides, Fasting, High | 150 to 300 | >300 to 500 | >500 to <1,000 | >1,000 |
| | 1.71 to 3.42 | >3.42 to 5.7 | >5.7 to 11.4 | >11.4 |
| <b>Magnesium</b> <sup>14</sup> , <b>Low</b> (mEq/L; <i>mmol/L</i> ) | 1.2 to <1.4 | 0.9 to <1.2 | 0.6 to <0.9 | <0.6 |
| | 0.60 to <0.70 | 0.45 to <0.60 | 0.30 to <0.45 | <0.30 |
| <b>Phosphate, Low</b> (mg/dL; mmol/L) | 2.0 to <lln< td=""><td>1.4 to &lt;2.0</td><td>1.0 to &lt;1.4</td><td>&lt;1.0</td></lln<> | 1.4 to <2.0 | 1.0 to <1.4 | <1.0 |
| | 0.65 to <lln< td=""><td>0.45 to &lt;0.65</td><td>0.32 to &lt;0.45</td><td>&lt;0.32</td></lln<> | 0.45 to <0.65 | 0.32 to <0.45 | <0.32 |
| <b>Potassium, High</b> (mEq/L; <i>mmol/L</i> ) | 5.6 to <6.0 | 6.0 to <6.5 | 6.5 to <7.0 | ≥7.0 |
| | 5.6 to <6.0 | 6.0 to <6.5 | 6.5 to <7.0 | ≥7.0 |
| <b>Potassium, Low</b> (mEq/L; <i>mmol/L</i> ) | 3.0 to <3.4 | 2.5 to <3.0 | 2.0 to <2.5 | <2.0 |
| | 3.0 to <3.4 | 2.5 to <3.0 | 2.0 to <2.5 | <2.0 |
| <b>Sodium, High</b> (mEq/L; mmol/L) | 146 to <150 | 150 to <154 | 154 to <160 | ≥160 |
| | 146 to <150 | 150 to <154 | 154 to <160 | ≥160 |
| <b>Sodium, Low</b> (mEq/L; <i>mmol/L</i> ) | 130 to <135 | 125 to <130 | 121 to <125 | ≤120 |
| | 130 to <135 | 125 to <130 | 121 to <125 | ≤ <i>1</i> 20 |
| Uric Acid, High (mg/dL; mmol/L) | 7.5 to <10.0 | 10.0 to <12.0 | 12.0 to <15.0 | ≥15.0 |
| | 0.45 to <0.59 | 0.59 to <0.71 | 0.71 to <0.89 | ≥0.89 |

<sup>\*</sup>Reminder: Choose the method that selects for the higher grade.

<sup>\*</sup>Reminder: An asymptomatic abnormal laboratory finding without an accompanying adverse event should not be reported to DAIDS in an expedited time frame unless it meets protocol-specific reporting requirements.

<sup>13</sup> Use the applicable formula (i.e., Cockcroft-Gault in mL/min or Schwartz, MDRD, CKD-Epi in mL/min/1.73m<sup>2</sup>). Sites should choose the method defined in their study and when not specified, use the method most relevant to the study population.

<sup>14</sup> To convert a magnesium value from mg/dL to mmol/L, laboratories should multiply by 0.4114.

| | | | _ | |
|----|-----|------|-----|----|
| 11 | ema | -4- | ۱., | ~ |
| ш | emz | 4110 | HO) | υv |

| Tiematology | | | | Conda 4 Datastialla |
|---|---|---|---|---|
| Parameter | Grade 1 Mild | Grade 2 Moderate | Grade 3 Severe | Grade 4 Potentially Life- Threatening |
| Absolute CD4+ Count,<br>Low (cell/mm³; cells/L)<br>(not HIV infected) | 300 to <400<br>300 to <400 | 200 to <300<br>200 to <300 | 100 to <200<br>100 to <200 | <100<br><100 |
| Absolute Lymphocyte Count, Low (cell/mm³; cells/L) (not HIV infected) | 600 to <650<br>0.600×10 <sup>9</sup> to<br><0.650×10 <sup>9</sup> | 500 to <600<br>0.500×10 <sup>9</sup> to<br><0.600×10 <sup>9</sup> | 350 to <500<br>0.350×10 <sup>9</sup> to<br><0.500×10 <sup>9</sup> | <350<br><0.350×10 <sup>9</sup> |
| Absolute Neutrophil<br>Count (ANC), Low<br>(cells/mm³; cells/L) | 800 to 1,000<br>0.800×10 <sup>9</sup> to 1.000×10 <sup>9</sup> | 600 to 799<br>0.600×10 <sup>9</sup> to 0.799×10 <sup>9</sup> | 400 to 599<br>0.400×10 <sup>9</sup> to 0.599×10 <sup>9</sup> | <400<br><0.400×10° |
| <b>Fibrinogen, Decreased</b> (mg/dL; <i>g/L</i> ) | 100 to <200<br>1.00 to <2.00 OR 0.75<br>to <1.00×LLN | 75 to <100<br>0.75 to <1.00 OR ≥0.50<br>to <0.75×LLN | 50 to <75<br>0.50 to <0.75 OR 0.25<br>to <0.50×LLN | <50<br><0.50 OR <0.25×LLN<br>OR Associated with<br>gross bleeding |
| Hemoglobin <sup>15</sup> , Low<br>(g/dL; mmol/L) <sup>16</sup><br>Male only | 10.0 to 10.9<br>6.19 to 6.76 | 9.0 to <10.0<br>5.57 to <6.19 | 7.0 to <9.0<br>4.34 to <5.57 | <7.0<br><4.34 |
| Hemoglobin <sup>15</sup> , Low (g/dL; mmol/L) <sup>16</sup> female only | 9.5 to 10.4<br>5.88 to 6.48 | 8.5 to <9.5<br>5.25 to <5.88 | 6.5 to <8.5<br>4.03 to <5.25 | <6.5<br><4.03 |
| INR, High (not on anticoagulation therapy) | 1.1 to <1.5×ULN | 1.5 to <2.0×ULN | 2.0 to <3.0×ULN | ≥3.0×ULN |
| Methemoglobin<br>(% hemoglobin) | 5.0 to <10.0% | 10.0 to <15.0% | 15.0 to <20.0% | ≥20.0% |
| PTT, High (not on anticoagulation therapy) | 1.1 to <1.66×ULN | 1.66 to <2.33×ULN | 2.33 to <3.00×ULN | ≥3.00×ULN |
| Platelets, Decreased (cells/mm³; cells/L) | 100,000 to <125,000<br>100.000×10 <sup>9</sup> to<br><125.000×10 <sup>9</sup> | 50,000 to <100,000<br>50.000×10 <sup>9</sup> to<br><100.000×10 <sup>9</sup> | 25,000 to <50,000<br>25.000×10 <sup>9</sup> to<br><50.000×10 <sup>9</sup> | <25,000<br><25.000×10 <sup>9</sup> |
| PT, High<br>(not on anticoagulation<br>therapy) | 1.1 to <1.25×ULN | 1.25 to <1.50×ULN | 1.50 to <3.00×ULN | ≥3.00×ULN |
| WBC, Decreased (cells/mm <sup>3</sup> ; <i>cells/L</i> ) | 2,000 to 2,499<br>2.000×10 <sup>9</sup> to 2.499×10 <sup>9</sup> | 1,500 to 1,999<br>1.500×10 <sup>9</sup> to 1.999×10 <sup>9</sup> | 1,000 to 1,499<br>1.000×10 <sup>9</sup> to 1.499×10 <sup>9</sup> | <1,000<br><1.000×10 <sup>9</sup> |

<sup>15</sup> Male and female sex are defined as sex at birth. For transgender participants who have been on hormone therapy for more than 6 consecutive months, grade hemoglobin based on the gender with which they identify (i.e., a transgender female should be graded using the female sex at birth hemoglobin laboratory values).

<sup>16</sup> The most commonly used conversion factor to convert g/dL to mmol/L is 0.6206. For grading hemoglobin results obtained by an analytic method with a conversion factor other than 0.6206, the result must be converted to g/dL using appropriate conversion factor for the particular laboratory.

# Urinalysis

| Parameter | Grade 1 Mild | Grade 2 Moderate | Grade 3 Severe | Grade 4 Potentially<br>Life- Threatening |
|---|---|---|---|---|
| Glycosuria (random collection tested by dipstick) | Trace to 1+ or ≤250 mg | 2+ or >250 to ≤500 mg | >2+ or >500 mg | NA |
| Hematuria (not to be<br>reported based on<br>dipstick findings or on<br>blood believed to be of<br>menstrual origin) | 6 to <10 RBCs per high<br>power field | ≥10 RBCs per high<br>power field | Gross, with or without<br>clots OR With RBC<br>casts OR Intervention<br>indicated | Life-threatening consequences |
| Proteinuria (random collection tested by dipstick) | 1+ | 2+ | 3+ or higher | NA |

#### 19.3 APPENDIX III – Cytochrome P450 2B6, 2C8, 2C9, and 2D6 Substrates

The following drugs are known substrates of CYP 2B6, 2C8, 2C9, and 2D6 and should be avoided while on treatment:

- 2B6: Artemisinin, bupropion, cyclophosphamide, efavirenz, ifosphamide, ketamine, meperidine, methadone, nevirapine, propafol
- 2C8: Amodiaquine, cerivastatin, paclitaxel, repaglinide, sorafenib, torsemide
- 2C9: NSAIDs: Diclofenac, ibuprofen, lornoxicam, meloxicam, naproxen, piroxicam, suprofen Oral Hypoglycemic Agents: Tolbutamide, glipizide Angiotensin II Blockers: Losartan, Irbesartan

Sulfonylureas: Glyburide, glibenclamide, glipizide, glimepiride, tolbutamide Other: Amitriptyline, celecoxib, fluoxetine, fluvastatin, glyburide, nateglinide, phenytoin-4-OH2, rosiglitazone, tamoxifen

• 2D6: Tamoxifen

Beta Blockers: Carvedilol, S-metoprolol, propafenone, timolol Antidepressants: Amitriptyline, clomipramine, desipramine, fluoxetine, imipramine, paroxetine, venlafaxine

Antipsychotics: Haloperidol, perphenazine, risperidone→9-OH, thioridazine, zuclopenthixol

Other: Alprenolol, amphetamine, aripiprazole, atomoxetine, bufuralol, chlorpheniramine, chlorpromazine, clonidine, codeine, debrisoquine, dexfenfluramine, dextromethorphan, donepezil, duloxetine, encainide, flecainide, fluvoxamine, lidocaine, metoclopramide, methoxyamphetamine, mexiletine, minaprine, nebivolol, nortriptyline, ondansetron, oxycodone, perhexiline, phenacetin, phenformin, promethazine, propafenone, propranolol, risperidone, sparteine, tramadol

Source: The Flockhart Table. http://medicine.iupui.edu/clinpharm/ddis/main-table# [Accessed 26 Apr 2018]